Protocol HPTN 083 Statistical Analysis Plan

# STATISTICAL ANALYSIS PLAN

# **Protocol HPTN 083**

A Phase 2b/3 Double Blind Safety and Efficacy Study of Injectable Cabotegravir Compared to Daily Oral Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC), For Pre-Exposure Prophylaxis in HIV-Uninfected Cisgender Men and Transgender Women who have Sex with Men

Effective Date: Effective on the date of final approval signature

Version 4.0

Prepared by

# Deborah Donnell HPTN SDMC Blinded Statistician

# STATISTICAL ANALYSIS PLAN

| Protocol Name: | A Phase 2b/3 Double Blind Safety and Efficacy Study of Injectable Cabotegravir Compared to Daily Oral Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC), For Pre-Exposure Prophylaxis in HIV-Uninfected Cisgender Men and Transgender Women who have Sex with Men |
|---|---|
| Protocol Number: | HPTN 083 |
| First version authors: | Deborah Donnell, Blinded Statistician |
| | Brett Hanscom, Unblinded Statistician |
| | Raphael Landovitz, HPTN 083 Protocol Chair |
| | Beatriz Grinsztejn, HPTN 083 Protocol Co-chair |
| Version: | 4.0 |


HPTN 083 Statistical Analysis Plan

| Author(s): | | |
|----------------------------------|-----------|-------|
| Deborah Donnell | | |
| Blinded Protocol<br>Statistician | Signature | Date: |
| Approvals: | | |
| NIAID Statistical Reviewer | Signature | Date: |


# **Table of Contents**

| ABB | REVIATI | ON AND DEFINITIONS | 5 |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 6 |
| 2. | STUD | Y OBJECTIVES GENERAL DESIGN CONSIDERATIONS | 6 |
| 1. | 2.1 | Purpose | 6 |
| | 2.2 | Design | 6 |
| | 2.3 | Population | 6 |
| | 2.4 | Study Size | 6 |
| | 2.5 | Study Duration | 6 |
| | 2.6 | Study Regimen and Follow-up | 7 |
| 3. | STUD | Y OBJECTIVES | 8 |
| | 3.2 | Secondary Objectives | 8 |
| | 3.3 | Tertiary Objectives | 8 |
| | 3.4 | Exploratory Objectives | 9 |
| 4. | STAT | ISTICAL CONSIDERATIONS | 9 |
| | 4.1 | Randomization | 9 |
| | 4.2 | Blinding | |
| | 4.3 | Sample size and Power | 10 |
| 5. | BLINI | DED REVIEW OF HIV ENDPOINTS AND PROTOCOL VIOLATIONS | 11 |
| | 5.1 | Blinded determination of HIV endpoints. | 11 |
| | 5.2 | Classification of protocol deviations | 11 |
| 6. | ANAL | YSIS POPULATIONS | 12 |
| | 6.1 | Intent to Treat (ITT) Population | |
| | 6.2 | Modified ITT (mITT) Population (Primary Efficacy) | |
| | 6.3 | Per-Protocol (PP) Population | |
| | 6.4 | Injection (Step 2) Efficacy Population | 13 |
| | 6.5 | Step 3 Population | 13 |
| | 6.6 | Safety Population (Primary Safety) | |
| | 6.7 | Injection Step 2 Safety Population | |
| | 6.8 | Longitudinal Pharmacokinetic CAB Concentration Population | |
| | 6.9 | TDF-FTC Adherence Population | |
| | 6.10 | Seroconverter Population | |
| | 6.11 | Primary Seroconverter Population | |
| | 6.12 | Enrollment Seroconverter Population | |
| | 6.13 | Subgroups | 14 |

Statistical Analysis Plan


HPTN 083 Statistical Analysis Plan

| 7. | STATI | STICAL ANALYSES | 14 |
|---|---|---|---|
| | 7.1 | General analysis considerations | 14 |
| | 7.2 | Interim Analyses and Data Monitoring Committee | 14 |
| | 7.3 | Efficacy Analyses | 16 |
| | 7.4 | Safety Analyses | 19 |
| | 7.5 | Secondary Analyses | 22 |
| 8. | MISSI | NG DATA AND IMPUTATIONS | 26 |
| | 8.1 | Missing Start and Stop Dates for Prior and Concomitant Medication, and Medical His | |
| | 8.2 | Missing Start and Stop Dates for Adverse Events | _ |
| 9. | MONI | TORING REPORTS | 28 |
| | 9.1 | Performance Metric Reports | 28 |
| | 9.2 | SMC Reports | 28 |
| | 9.3 | DSMB Reports | 28 |
| | 9.4 | Clinical Study Report | 29 |
| 10. | REVIS | IONS OF THE SAP | 30 |
| | 10.1. | Changes in version 2.0 of the SAP | 30 |
| | 10.2 | Changes in version 3.0 of the SAP | 31 |
| | 10.3 | Changes in version 4.0 of the SAP | 32 |
| CHAN | NGE HIS | TORY | 33 |
| REFE | RENCES | S | 33 |
| APPE | NDIX A | VISIT WINDOWS | 35 |
| APPE | NDIX B | DEFINITION OF SUBGROUPS | 37 |
| APPE | NDIX C | DETAILS OF EFFICACY ANALYSIS DEFINITIONS | 38 |
| APPE | NDIX D | STUDY DRUG DISCONTINUATION ANALYSIS DUE TO SAFETY | 40 |
| APPE | NDIX E | DEFINITIONS OF REGIONS FOR STUDY SITES | 41 |
| APPE | NDIX F: | ADVERSE EVENTS OF SPECIAL INTEREST | 42 |

# **ABBREVIATION AND DEFINITIONS**

| ALT | Alanine Aminotransferase |
|---------|---------------------------------------------|
| ARV | Antiretroviral |
| AST | Aspartate Aminotransferase |
| CAB | Cabotegravir |
| CI | Confidence Interval |
| Cr | Creatinine Clearance |
| CRF | Case Report Form |
| csHT | cross-sex Hormone Therapy |
| DBS | Dried Blood Spots |
| DSMB | Data Safety Monitoring Board |
| ECG | Electrocardiogram |
| ехр | Exponential |
| GFR | Glomerular Filtration Rate |
| HBsAg+ | Hepatitis B surface Antigen |
| HCV | Hepatitis C Virus |
| HIV | Human Immunodeficiency Virus |
| HR | Hazard Ratio |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation |
| IDU | Injection drug user |
| IM | Intramuscular |
| loR | Investigator of Record |
| ITT | Intent to Treat |
| LFT | Liver Function Test |
| MSM | Men who have Sex with Men |
| NI | Non-Inferiority |
| OBSP | On Blinded Study Product |
| PEP | Post-Exposure Prophylaxis |
| PrEP | Pre-Exposure Prophylaxis |
| PT | Preferred Term |
| RR | Relative Risk |
| SAP | Statistical Analysis Plan |
| SDMC | Statistical and Data Management Center |
| SOC | System Organ Class |
| STD | Sexually Transmitted Disease |
| STIs | Sexually Transmitted Infections |
| TDF/FTC | Tenofovir Disoproxil Fumarate/Emtricitabine |
| TFV | Tenofovir |
| TFV-DP | Tenofovir Diphosphate |
| TGW | Transgender Women |


#### 1. INTRODUCTION

This statistical analysis plan (SAP) details the statistical procedures that address the primary study objectives specified in Version 3.0 of *Protocol HPTN 083: A Phase 2b/3 Double Blind Safety and Efficacy Study of Injectable Cabotegravir Compared to Daily Oral Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC), For Pre-Exposure Prophylaxis in HIV-Uninfected Cisgender Men and Transgender Women who have Sex with Men.* A brief description of secondary endpoint analyses is included. New versions of the SAP will be issued to document updates and changes in the plan. Any meaningful changes or additions to this SAP (e.g., in response to protocol amendments or violations of assumptions underlying pre-planned analyses), and the timing of such changes in relation to unblinding of statisticians performing the analyses, will be documented in a designated section of the SAP. Analysis plans for sub-studies not addressed in the protocol, and for secondary analyses not anticipated prior to study completion, and for exploratory analyses will be developed as separate documents.

Plans for formal interim analysis of trial data are outlined in Section 7.2. A more detailed plan is documented separately in HPTN 083 Interim Monitoring Guidelines. Any substantive modifications to analysis methods or type I error control made in response to DSMB reviews or changes in the protocol will be documented in subsequent versions of the SAP. In DSMB reviews, the HPTN Statistical and Data Management Center (SDMC) will routinely report on operational metrics (e.g., rates of recruitment, retention, study drug discontinuation). These reports are also routinely shared with the study sites to monitor operational performance based on these metrics. No aggregate reporting of HIV infection events or safety data are included in these routine reports to study sites, the format and schedule of which are not considered further in this SAP.

#### 2. STUDY OBJECTIVES GENERAL DESIGN CONSIDERATIONS

#### 2.1 Purpose

The purpose of this study is to evaluate the safety and efficacy of the injectable agent, cabotegravir (CAB LA), for pre-exposure prophylaxis (PrEP) in HIV-uninfected cisgender men and transgender women who have sex with men (MSM and TGW).

#### 2.2 Design

Multi-site, double blind, two-arm, randomized (1:1), controlled non-inferiority trial of the efficacy of CAB LA compared to daily oral tenofovir disoproxyl fumarate (TDF)/emtricitabine (FTC) for HIV prevention.

### 2.3 Population

HIV-uninfected MSM and TGW at risk for acquiring HIV infection, ages 18 or older.

#### 2.4 Study Size

Approximately 5000, 2500 per arm. Following DSMB review in November 2019 the sample size was increased from 4500 to 5000, as documented in the DSMB recommendations.

# 2.5 Study Duration

Approximately 5.5 years total, with individual participants being followed between 2.5 years (for the latest enrolling participants) to 4 years (for the earliest enrolling participants). Accrual will require approximately 130 weeks. In Step 1, participants will


receive oral tablets for 5 weeks. In Step 2, participants will receive injections (as a single injection at two time points 4 weeks apart and every 8 weeks thereafter) and daily oral tablets. Step 2 will be continued until the required number endpoints is reached, or the maximum number of person years specified in the protocol is reached, whichever occurs first. Participants will all be simultaneously unblinded at the conclusion of Step 2. In Step 3, all participants on blinded study drug will receive open-label daily oral TDF/FTC for up to 48 weeks. Participants will therefore be followed for a maximum of four years, including up to three years on blinded study medication and 48 weeks on open-label daily oral TDF/FTC. All participants will be transitioned to locally-available HIV prevention services, including services for PrEP, if available, at the end of their participation in the study.

#### 2.6 Study Regimen and Follow-up

Once randomized to one of two arms, participants will move through the following steps (active drugs are shown in bold text):

#### Step 1:

Arm A – **Daily oral CAB** (30 mg tablets) and oral TDF/FTC placebo for five weeks

Arm B – **Daily oral TDF/FTC** (300 mg/200 mg fixed-dose combination tablets) and oral CAB placebo for five weeks

A participant that becomes HIV-infected during Step 1 of the study will permanently discontinue study product, be terminated from the study, and referred for HIV-related care. Individuals who discontinue study participation after receiving oral product in Step 1, but do not receive any study product in Step 2 will be followed annually with HIV testing for a maximum of three years from enrollment.

# Step 2:

Arm A – **CAB LA** (600 mg as a single intramuscular [IM] injection at two time points 4 weeks apart and every 8 weeks thereafter) and daily oral TDF/FTC placebo.

Arm B – **Daily oral TDF/FTC** (300/200 mg fixed-dose combination tablets) and IM placebo at two time points 4 weeks apart and every 8 weeks thereafter (matching vehicle, identical volume as active injectable product in Arm A).

For individual participants 8 weekly injections/pills will continue until three years of follow-up is complete, to Week 153, with the last injection provided and the last blinded oral study product dispensed at Week 145. Participants who prematurely discontinue blinded study products during Step 2 (having received at least one injection) for any reason other than HIV infection will transition to Step 3 early.

This step will continue until (a) the maximum number of endpoints have been observed or (b) the maximum number of person years specified in the protocol is observed, whichever occurs first.

A participant who becomes HIV-infected during Step 2 of the study will permanently discontinue study product, be placed on immediate suppressive ART, and will be followed at quarterly intervals for 52 weeks after their last injection prior to diagnosis of HIV in order to test for safety parameters, as well


as CD4 cell count and HIV viral load. After 52 weeks, they will be terminated from the study and transitioned to continued HIV-related care.

# Step 3:

Both arms: **Open-label daily oral TDF/FTC** no later than 8 weeks after the last injection (in order to provide ongoing HIV prophylactic coverage to high risk individuals), for up to 48 weeks. Participants will then transition to locally-available HIV prevention services, including services for PrEP, if available. A participant with confirmed HIV infection during Step 3 will be followed at least for the duration of Step 3, with possible additional assessments and follow-up to be determined by the Clinical Management Committee (CMC).

# 3. Study Objectives

### 3.1 Primary Objectives

- To compare HIV incidence among participants randomized to oral CAB/CAB LA (oral lead in and injections) vs. oral TDF/FTC (Steps 1 and 2)
- To compare the safety of oral CAB/CAB LA vs. oral TDF/FTC

# 3.2 Secondary Objectives

- To compare HIV incidence among participants receiving CAB LA injections vs. oral TDF/FTC in Step 2
- To compare HIV incidence among participants receiving CAB LA injections vs. oral TDF/FTC (Steps 1, 2, and 3 combined)
- To compare HIV incidence among participants randomized to CAB LA injections vs. oral TDF/FTC while taking open label TDF/FTC (Step 3 only, descriptive)
- To compare the change in risk of HIV acquisition between CAB and oral TDF/FTC strategies (Arm A and Arm B) as participants progress from Step 2 to Step 3 (i.e. post week 153)
- To compare HIV incidence among the subgroups of participants receiving oral CAB/CAB LA vs. oral TDF/FTC by region, age, race, ethnicity, baseline risk, and gender identity
- To compare changes in renal function, liver function, and bone mineral density (BMD) among participants receiving oral CAB/CAB LA vs. oral TDF/FTC
- To evaluate and compare rates of HIV drug resistance among participants who acquire HIV infection during the study among participants receiving oral CAB/CAB LA vs oral TDF/FTC
- To compare the acceptability of and preferences for CAB LA vs. oral TDF/FTC
- To compare changes in weight, blood pressure, and pulse, fasting glucose, and fasting lipids among participants receiving oral CAB/CAB LA vs. oral TDF/FTC

# 3.3 Tertiary Objectives

To examine the association between levels of adherence and HIV incidence


- To compare and describe the rates, patterns, and correlates of adherence to CAB LA vs oral TDF/FTC, in aggregate and by psychosocial/demographic variables
- To estimate changes in sexual-risk behavior as measured by self-report and rates of incident gonorrhea, chlamydia, and syphilis in the study population
- To compare the resource utilization and programmatic costs of long-acting injectable PrEP vs. daily oral PrEP vs. no PrEP for HIV uninfected MSM and TGW in the US, Brazil, South Africa
- To use mathematical simulation to project the short- and long-term clinical impact, cost projections, budgetary impact, and incremental cost-effectiveness of long-acting injectable PrEP vs. daily oral PrEP vs. no PrEP for HIV uninfected MSM and TGW in the US, Brazil, South Africa

#### 3.4 Exploratory Objectives

- To perform secondary laboratory assessments that may include evaluation of factors related to HIV infection, hepatitis infection, or sexually transmitted infections (STIs); antiretroviral (ARV) drug use; pharmacogenomics; characterization of HIV in infected participants; and evaluation of laboratory assays related to the study objectives
- To explore possible drug-drug interactions between cross-sex hormone therapy (csHT) and cabotegravir and TDF/FTC in a subset of TGW taking commonly prescribed cross-sex hormone therapy regimens

#### 4. STATISTICAL CONSIDERATIONS

#### 4.1 Randomization

Enrolled participants will be randomized to one of two study arms in a 1:1 ratio. Randomization will be stratified by study site, and a permuted blocks design will be used to ensure balanced treatment assignments within study site. Once a participant has been enrolled, the random-arm assignment will be automatically retrieved from the central server and provided to site pharmacist via the *Balance* module in the *Medidata Rave* web interface. Only the pharmacist will know which oral and injectable products are being dispensed.

#### 4.2 Blinding

In this double-blind double-dummy design, both oral and injectable study products are blinded, and both oral and injectable products are administered to each participant.

Step 1: Blinded oral products

Arm A: Oral CAB tablets 30 mg, one tablet orally daily for five weeks, with or without food AND placebo for TDF/FTC tablets, one tablet orally daily for 5 weeks, with or without food

Arm B: TDF/FTC 300 mg/200 mg fixed dose combination tablet, one tablet orally daily for five weeks, with or without food AND placebo for oral CAB tablet, orally daily for 5 weeks, with or without food

Step 2 – Blinded injections and blinded daily oral pills:


Arm A: CAB LA 600 mg administered as one 3 mL (600 mg) intramuscular IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter, AND placebo for TDF/FTC tablet, one tablet orally daily with or without food

Arm B: TDF/FTC 300 mg/200 mg fixed dost combination tablet, one tablet orally daily, with or without food AND placebo for CAB LA (Intralipid 20% fat emulsion infusion) administered as one 3mL intramuscular (IM) injection in the gluteal muscle as two time points 4 weeks apart and every 8 weeks thereafter

Study site staff and participants will be blinded to the random assignments, with the exception of the site Pharmacist of Record or their designee. Blinding will be maintained until the trial is completed or stopped, i.e., the trial is stopped early, or the required number of endpoints or person years has been met (with the exception of emergency unblinding). At a specified time directed by the HPTN SDMC, participants will be notified of their treatment assignment. In addition, as noted in Section 5.14.2, an Investigator can request unblinding to the HPTN SDMC in the event that a participant becomes infected with HIV during the study, and the SDMC will assist in directly providing the participant's primary health care provider the randomized arm assignment information per their SOP; the randomized assignment will not be provided to the site where the participant was enrolled and followed.

If, in the judgment of the site investigator of record (IoR), or in the judgment of the participant's medical provider and the site IoR, a medical event is of sufficient extreme severity that it requires the immediate unblinding of a participant, the site IoR may proceed with unblinding a participant. Emergency unblinding is expected to be extremely rare. It should only occur in the setting of a potentially life-threatening clinical event, and if knowing the participant's treatment assignment would affect decisions regarding the participant's immediate medical management. Both conditions must be satisfied. Study site pharmacists who prepare the study drugs are not blinded.

#### 4.3 Sample size and Power

The sample size was computed assuming CAB LA is 25% more effective than TDF/FTC, for a non-inferiority margin of 1.23. Approximately 172 observed HIV-infections will provide 90% power to rule out a non-inferiority margin of HR=1.23, with one-sided type-I error alpha = 0.025. This non-inferiority margin is an M2 margin based on an inversevariance weighted meta-analysis of three randomized controlled trials of TDF/FTC versus placebo in MSM: iPrex, iPERGAY, and PROUD(1-3). The M2 margin is defined as the reduced bound that is designed to preserve a clinically acceptable amount of the benefit provided by the active control (TDF/FTC). Setting M2 to be 50% of M1 (on the log scale in the case of hazard ratios) is considered to be conservative. M1 is defined as the lower limit of the 95% confidence interval around the placebo versus active-control HR estimate (1.51, based on the meta-analysis). Once the stated number of HIV-infections have been observed, non-inferiority will be established if the estimated CAB LA versus TDF/FTC hazard ratio point estimate is approximately 0.90 or less (indicating a 10% advantage of CAB LA over TDF/FTC), and superiority will be established if the hazard ratio point estimate is approximately 0.74 or less (indicating a 26% advantage of CAB LA over TDF/FTC). The power to detect superiority is 47%. Sample size was computed using RCTDesign package in R and confirmed in nQuery.


#### 5. BLINDED REVIEW OF HIV ENDPOINTS AND PROTOCOL VIOLATIONS

#### 5.1 Blinded determination of HIV endpoints.

A blinded special endpoint adjudication committee (SEAC) is responsible for determining the HIV primary endpoints of the study, i.e. HIV infections occurring after enrollment and during primary analysis follow-up

Prior to each DSMB interim monitoring efficacy review, and prior to unblinding of the final analysis,), the SEAC will engage in a blinded review of all cases with positive/reactive HIV test results to adjudicate study endpoints. The review will make blinded decisions about the confirmation and timing of HIV infection and adjudicate any unexpected issues in the data affecting the primary efficacy endpoints. Data, algorithms and processes for SEAC review are documented in *Terms of reference for HPTN 083 SEAC* and summarized here.

Site testing typically first identifies participants with a reactive HIV test. The HPTN 083 seroconverter alias assist the site in managing the care of potential seroconverters, including additional testing, study drug hold etc. Subsequent testing at the LC, incorporating results from visits before, at and after visits with a reactive test are used to confirm HIV status of each participant with a reactive test.

Endpoint review will make final decisions on all cases of HIV acquisition and data related to the timing of HIV infection. Particular attention will be focused on the following:

- 1. All cases designated as infected at enrollment.
- 2. All cases where infection occurred at a visit prior to detection of infection by the site. In particular, this would include review of infections first detected in Step 3 that are subsequently determined to have occurred in Step 2.
- 3. All cases where site testing did not follow the HIV testing algorithm for determining infection for any reason.
- 4. Any other unusual cases determined by the LC, stat center or seroconverter alias.

#### 5.2 Classification of protocol deviations

All protocol deviations will be reported and reviewed on a regular basis, and each case will be managed clinically and with regard to ongoing product administration by the CMC and DAIDS MOs during the course of the trial. Certain serious protocol deviations, identified during the blinded review, may warrant the exclusion of participants from the mITT and/or Per-Protocol analysis. Generally, exclusions from the mITT analysis are expected to be limited to participants deemed inappropriately enrolled and resulting in termination from the study. Any exclusion must be carefully adjudicated and scientifically justified prior to breaking the blind. The following list may be updated to reflect unanticipated protocol violations at the time of blinded review.

**Protocol Violations** 

Potentially exclusionary from ITT analyses:

Under 18 at enrollment Not male at birth IDU at enrollment ICF violations


#### Potentially exclusionary from the per-protocol analyses:

HCV positive at enrollment

Lab abnormality or relevant medical condition at enrollment

Prior participation in HIV vaccine trial

Incorrect study product received\*

Prohibited concomitant medicine use\*

**Buttock implant\*** 

Did not meet sexual risk criteria

HBsAa+

History of liver disease

Coagulopathy

Allergy to components

History of seizure

Missed HIV testing elements

Missed safety elements (e.g., LFTs, Cr)

Incorrect/inappropriate amount of study product dispensed\*

Inadequate adherence for progression to step 2

Injection administration/product dispensation prior to appropriate lab results available\*

Outside protocol TDF/FTC use during protocol (outside PEP)\*

\*Potential partial exclusion. Exclude (censor) from analyses at the time of the deviation

# Minor – not exclusionary:

Co-enrollment in another study without permission

Clinically significant CV disease

Inflammatory skin condition without CMC approval

Tattoo on buttock without CMC approval

Visits out of window without with/without CMC approval

Missed labs/assessments on-study (except HIV testing, LFTs, Cr)

Non-fasting lipids

Missed STD testing

Missed/incorrect f/u for laboratory or clinical AEs

ECG parameter violations

#### 6. ANALYSIS POPULATIONS

#### 6.1 Intent to Treat (ITT) Population

All participants who were randomized, excluding those who were inappropriately enrolled

#### 6.2 Modified ITT (mITT) Population (Primary Efficacy)

The ITT population, excluding those who were found to be HIV infected at randomization.

Analysis period: Primary analysis follow-up data will include study time through the completion of the blinded injection phase of study follow-up (i.e. Week 153 or the study-wide transition to


Step 3, or end of the blinded phase of the study, whichever occurs first). Inclusion/exclusion of visits are detailed in Appendix A.

### 6.3 Per-Protocol (PP) Population

The mITT population excluding all participants with protocol violations that were judged to be exclusionary from the per-protocol population.

### 6.4 Injection (Step 2) Efficacy Population

The mITT population who receive at least one injection and are uninfected at the time of the first injection.

Analysis period: Follow-up time will include primary analysis study time from the time of the first injection through the completion of the blinded injection phase of study follow-up.

# 6.5 Step 3 Population

All mITT participants who are uninfected at the start of Step 3 follow-up, (i.e. the Week 153/ study-wide transition to Step 3).

#### 6.6 Safety Population (Primary Safety)

All ITT participants who received any oral or injectable product. All safety events occurring on study will be reported.

Step 1 adverse events will include all adverse events occurring until the first injection date, or 120 days post randomization, whichever comes first.

### 6.7 Injection Step 2 Safety Population

All Safety Population participants who receive at least one injection.

Step 2 safety will include all adverse events occurring from the first injection date through 48 weeks after the last injection.

#### 6.8 Longitudinal Pharmacokinetic CAB Concentration Population

A longitudinal evaluation of CAB PK in the CAB arm will be conducted in 200 participants who received all injections up through week 57, selected with the following regional distribution

- 5% US sites Non-African American (10 participants)
- 5% US sites African American (10 participants)
- 40% Asia (80 participants; 50% TGW using gender affirming hormonal therapy/cross-sex hormonal therapy)
- 40% Latin America (80 participants, 50% TGW using gender affirming hormonal therapy/cross-sex hormonal therapy)
- 10% Africa (20 participants)

This population will be used for the CAB concentration listing and to enhance the population represented in the global modelling of CAB-LA PK.

# 6.9 TDF-FTC Adherence Population

Cohort of approximately 400 participants randomly selected at baseline from the oral TDF/FTC arm.

#### 6.10 Seroconverter Population

All ITT participants who are identified to be HIV infected following randomization.


#### 6.11 Primary Seroconverter Population

All ITT participants who are HIV-uninfected at randomization and acquire HIV infection during primary analysis follow-up.

# **6.12 Enrollment Seroconverter Population**

All ITT participants who were determined to be HIV-infected at randomization

### 6.13 Subgroups

Important participant subgroups are

- Region: USA, Latin America, Asia, Africa
- Age:<30 vs ≥30 years old</li>
- Race/Ethnicity: US Black vs non-Black; Hispanic (Yes/No)
- Baseline risk:
  - ≤/> median number of sexual partners
  - ≤/> median report of condomless receptive anal sex
- Gender identity: MSM/TGW.
- Detailed definitions of subgroups are given in Appendix B

#### 7. STATISTICAL ANALYSES

#### 7.1 General analysis considerations

#### **Summary statistics**

Summary statistics for categorical variables will include frequency and percentage. For continuous variables, number of subjects with non-missing value (n), mean, median, Q1, Q3, standard deviation (SD), minimum (min), and maximum (max) will be reported. Baseline is defined as Visit 2.0 (Enrollment). All summaries and analyses will be presented by treatment group. Any deviations from the original statistical plan will be described in the final report.

#### **Visit Windows**

All data will be tabulated per the evaluation visit as recorded on the CRF even if the assessment is outside of the visit window. In data listings, the relative day, of all dates will be presented e.g. from date of randomization, or date of last injection.

#### 7.2 Interim Analyses and Data Monitoring Committee

A summary of the planned approach to interim monitoring is given here. Detailed guidance for early stopping is contained in a separate document: HPTN 083 Monitoring Guidelines.

#### 7.2.1 Interim Monitoring of drug levels

Population: TDF/FTC Adherence Population


Plasma and DBS samples from the TDF/FTC ADHERENCE cohort will be assessed for TFV and TFV-DP concentrations throughout the trial. These data will not be available to the protocol team. Data on TDF/FTC adherence, as measured by plasma and DBS concentrations, will be presented to the DSMB in each DSMB report. This will allow the DSMB to monitor the adherence to oral PrEP and assess the likelihood of reduced HIV acquisition in the TDF/FTC arm. In the event the TDF/FTC adherence appears to be substantially lower than assumed in the protocol, the DSMB can evaluate potential communication with the protocol team leadership if it is thought that actions could be taken to improve adherence to the daily oral medication. The detectable plasma concentrations will be used to estimate the average adherence in the cohort and model, based on plasma concentration data reported from prior placebo randomized trials, the estimated efficacy of TDF/FTC in the cohort. Comparable efficacy data is not available for DBS, although data from DBS concentrations achieved in directly observed therapy studies will permit additional interpretation of the average adherence to TDF/FTC.

#### 7.2.1 Interim Endpoint Analyses

Formal interim statistical analyses are planned for three time points during the trial, with analysis times corresponding to approximately when ¼, ½ and ¾ of the estimated maximum number of HIV infections have been observed. Interim analysis results will be provided to the DSMB at the scheduled DSMB meeting immediately following the time each interim number of events have been observed, or at other time requested by the protocol team or DSMB. The DSMB will receive updated numbers of infections observed at each DSMB meeting.

### Population: mITT

Analysis: This analysis will mimic the first objective in the primary analysis with the exception that the interim estimated hazard ratio will be compared to the pre-specified group-sequential stopping boundaries instead of to the non-inferiority margin. It was initially planned to monitor the trial early for early stopping based on the interim monitoring boundary for superiority, or early evidence that oral CAB/CAB LA is definitively less effective than oral TDF/FTC. In light of the disruption to the dispensing of study drug caused by COVID-19 beginning in Mar 2020, the interim monitoring guidance was changed to recommend early stopping based on the non-inferiority boundary, i.e. to recommend stopping based on crossing the O'Brien-Fleming boundary for non-inferiority.

The primary endpoint will be time to detection of HIV infection (time from randomization to midpoint between last HIV negative and first detection). HIV infection status will be assumed to be negative at all missing visits, if any, prior to the first reactive/positive HIV test. In accordance with intention-to-treat principles all participants will be classified into the study arm to which they were randomized. For study participants who do not acquire HIV infection, study time will be censored at the most recent HIV test, as specified in Appendix C. Censoring will be treated as uninformative. A Cox-regression model will be used to estimate the hazard ratio comparing the risk of HIV infection in Arm A (oral CAB/CAB LA) to Arm B (TDF/FTC), and the estimated hazard ratio will be compared to the O'Brien Fleming boundaries for non-inferiority and harm. Boundaries will be estimated based on the faction of observed information calculated based on the planned study design of a maximum of 172 events.


### **ON BLINDED STUDY PRODUCT Analysis**

To support the non-inferiority hypothesis, a supportive analysis will be presented using the OBSP censoring in the Injection (Step 2) Efficacy population (see Section 7.3.4), where study follow-up is censored when a participant does not receive blinded injection study product on time.

# 7.3 Efficacy Analyses

### 7.3.1 Study Hypothesis

The statistical hypotheses being tested in this double-blind double-dummy non-inferiority trial are:

Ho: HR (CAB-LA vs FTC/TDF) = 1.23 Ha: HR (CAB-LA vs FTC/TDF) < 1.23

# 7.3.2 Primary Endpoint

The primary endpoint is HIV-infection occurring after study enrollment. (See Section 5.1) The time to HIV infection will be calculated as the time from randomization to the midpoint between first visit where HIV infection was present and the most recent prior visit where HIV infection was not detectable.

#### 7.3.3 Primary Analyses

Objective: To compare HIV incidence among participants randomized to oral CAB/CAB LA (oral lead in and injections) vs. oral TDF/FTC (Steps 1 and 2)

Population: mITT

Censoring time: Study time is censored at the completion of the blinded injection phase of study follow-up (i.e. Week 153 or the study-wide transition to Step 3, or end of the blinded phase of the study, whichever occurs first).

Descriptive analysis: The number of participants, number of infections and cumulative person years will be presented by arm and overall. Incidence rates in each group will be calculated as the number of HIV infections divided by the total observed person time. Confidence intervals will be computed assuming infections are distributed according to a Poisson distribution. A Kaplan Meier plot will be used to display the cumulative rates of acquired HIV-infections by arm (i.e. 1 – KM(t))). Cumulative incidence rates of HIV detection at 12, 24, and 36 months will be reported from the Kaplan Meier plot by study arm and overall, with 95% confidence intervals calculated from the pointwise standard errors, assuming an asymptotic Normal distribution. Participants who are randomized and receive study product but are later determined to have been infected at enrollment are not included in this analysis and will be reported separately.

Statistical Analysis: In accordance with intention-to-treat (ITT) principles all eligible participants not infected at enrollment are included, classified according to randomized study arm. The primary mITT population includes primary analysis time for participants who stop injections early and could have subsequently initiated open label TDF/FTC. Person time in primary analysis is the time from enrollment to the first of (a) midpoint of interval where HIV infection was detected, (b) the last HIV test included in the primary analysis period. For study participants who do not acquire HIV infection, study time will be censored at the last HIV test in primary analysis follow-up. Details of the censoring for


the primary analysis follow-up are in Appendix C. Censoring will be treated as uninformative.

A Cox-regression model, stratified by region, with study arm as the only covariate will be used to estimate HR<sub>ITT</sub>: the hazard ratio comparing the risk of HIV infection in Arm A (oral CAB/CAB LA) to Arm B (oral TDF/FTC) and generate the 95% Wald-based confidence interval. The upper bound of the 95% confidence interval will be compared to the pre-specified non-inferiority margin of 1.23, with an upper 95% confidence bound less than 1.23 indicating non-inferiority.

#### Interpretation of the primary ITT analysis when H₀ is not rejected

In a scenario where the primary ITT analysis just fails to show non-inferiority, that is, the upper confidence limit on the hazard ratio is larger than the NI margin by a small amount, consideration will be given to determining whether CAB LA may provide important levels of benefit as compared to placebo. According to the FDA guidance document on NI trials(4):

Failure to exclude inferiority relative to M1 means there is no assurance of any effect. Just as it would be unusual to accept a placebo-controlled study as positive (i.e., a finding of superiority) with p > 0.05, it would be unusual to accept an NI study as positive (i.e., a finding of non-inferiority) where the upper bound of the 95% confidence interval was > M1. On the other hand, failing to exclude M2 by a small amount may be acceptable, as the small amount would not suggest the absence of an effect of the drug.

Provided that adherence to TDF/FTC is approximately as expected (57.5%) or higher, if HR<sub>ITT</sub> is not shown to be conclusively less than the pre-defined (M2) margin 1.23, but clearly and definitively rules out the M1 margin (1.51), it may be appropriate to discuss whether the trial results are consistent with CAB LA providing clinically important protection superior to placebo.

# Recomputation of the NI margin when TDF/FTC adherence is lower or higher than assumed

Of key importance in a non-inferiority trial is the assumption that the active-control therapy (oral TDF/FTC in our case) will be as effective as it was in the prior trials used to construct the NI margin. This is referred to as the constancy assumption. Although it is impossible to know with certainty whether the constancy assumption is true, if there exist strong, measurable predictors of effectiveness it may be possible to determine the degree to which the constancy assumption is not true. In the case of oral TDF/FTC it has been shown that drug adherence is a powerful predictor of effectiveness. In order to assess adherence, a random sample of participants in the TDF/FTC arm (the "TDF/FTC Adherence Cohort", described below) will be selected for laboratory testing of drug levels in plasma. As per section 7.4 in the protocol, if observed adherence rates are substantially outside the range of what was projected for the trial, i.e. adherence is lower than 50% or higher than 65%, the NI margin will be recomputed based on the methods described by Hanscom et al. (2017), and used to help gauge the potential prevention efficacy of CAB LA. The recomputed margin will not replace the pre-specified primary analysis margin or change the conclusion of the primary analysis, but may provide valuable information with respect to determining the prevention effectiveness of CAB LA.

TDF/FTC Adherence Cohort: A sample of 400 participants in the active TDF/FTC arm will be selected at random during the enrollment period and available plasma samples from selected visits (weeks 4, 9, 33, 57, 81, 105, 129, 153, 177) will be assessed for the


presence of TDF/FTC and associated metabolites. The TDF/FTC adherence cohort will be selected to ensure uniform representation over the course of the enrollment period. Random selection of this cohort will be stratified by geographic region (Latin America, Asia, United States, and Africa), and proportionally representative. Average, study-wide adherence will be computed as the overall proportion of all tested samples where TFV is detected in plasma (i.e. concentrations greater than 0.31 ng/ml).

Adapted NI Margin: The adapted NI margin will be based on the estimated TDF/FTC effectiveness given the observed adherence to TDF/FTC in the study cohort. Adherence to TDF/FTC is assessed as the proportion of tested samples in the adherence cohort who have detectable TFV in plasma. This is estimated using the meta-analysis regression equation derived from all prior randomized placebo controlled trials of oral TDF/FTC (5):

Relative Risk (TDF/FTC vs Placebo) = exp(0.735 - 2.439 x adherence)

The corresponding lower 95% confidence limit for this estimated relative risk becomes the revised M1 margin, which we will refer to as M1\*. The adapted NI margin is then computed so as to assure that at least half of the observed TDF/FTC benefit is preserved by CAB, and in addition that the margin requires CAB to be at least 15% more effective than placebo. This is accomplished by setting the margin as follows:

Adapted NI Margin =  $Min(Sqrt(M1^*), 0.85 \times M1^*)$ ,

where Sqrt(M1\*) represents the point at which half of the observed TDF/FTC benefit is preserved, and 0.85 x M1\* represents a 15% improvement over placebo. Note that if TDF/FTC adherence is so low that M1\* is less than or equal to 1.17, the adapted NI margin will be less than 1.0, indicating that super superiority is required to assure that CAB is at least 15% more effective than placebo.

# 7.3.4 Supportive analyses of the primary efficacy results while on blinded study product

In a non-inferiority trial, where all participants are on active treatment, the ITT analysis can be anti-conservative if adherence to either regimen is poor. The efficacy analysis restricted to time while on blinded study product (OBSP) will be a supportive analysis conducted to verify consistency with the ITT analysis, and understand the potential mechanisms for lack of consistency if that occurs. If the ITT and OBSP results are discrepant, possible reasons for the discrepancy will be carefully explored. For example,

- 1) If the experimental therapy is as biologically effective as the active control, but adherence is low in the active control arm, the ITT analysis would likely show that the experimental therapy was superior to the control (HR<sub>ITT</sub> < 1.0, a non-conservative result), while the OBSP analysis would be expected to show equal effectiveness (HR<sub>OBSP</sub> = 1.0).
- 2) If the experimental drug is biologically inferior, and adherence to active control was low, the ITT relative effectiveness  $HR_{ITT}$  would be expected to be closer to 1 ( $HR_{ITT} < HR_{OBSP}$ ) than the OBSP relative effectiveness ( $HR_{OBSP} > 1.0$ ).
- 3) If the experimental drug is truly superior and active control arm adherence in the experimental arm was moderate, both analyses would be expected to show superiority, but the ITT effectiveness would be expected to be stronger than the OBSP analysis (HR<sub>ITT</sub> < HR<sub>OBSP</sub> < 1.0).

It is worth noting that the expected differences between  $HR_{\text{ITT}}$  and  $HR_{\text{OBSP}}$  are quite different in this trial than in a typical non-interiority trial. In this trial the experimental


therapy is given by clinician-administered injection and therefore adherence is expected to be high. The active-control therapy, on the other hand, is given by self-administered oral tablets and hence adherence could be low. This could lead to substantial differences in adherence between treatment arms, which could lead to the results described above. In a typical non-inferiority trial both treatments are administered using the identical method, and hence any lack of adherence will affect both study arms equally. In general, this means that HR<sub>ITT</sub> is expected to be closer to 1.0 than HR<sub>OBSP</sub>, regardless of whether the experimental therapy is more or less effective than the active control.

Population: Injection Step 2 Efficacy population

Censoring time: For ON BLINDED STUDY PRODUCT (OBSP) analysis, study time is censored at the first time during the blinded injection phase of study follow-up when study injections are not received on the protocol schedule for any reason. Details of the OBSP censoring definitions are given in Appendix C.

Descriptive analysis: Same as the primary analysis, with participants, HIV infections and follow-up time restricted to the dataset.

Statistical Analysis:

The intent of this analysis is to assess relative effectiveness during the study time after randomization when the participant remained consistently on blinded injectable product. All participants who received an injection are included, with study time up to the first time the blinded injection is not given on time for any reason.

Censoring will be treated as uninformative. A Cox-regression model, stratified by region, with study arm as the only covariate will be used to estimate the hazard ratio comparing the risk of HIV infection in Arm A (oral CAB/CAB LA) to Arm B (oral TDF/FTC) and generate the 95% Wald-based confidence interval. The relative OBSP effectiveness, together with available lab-based assessments of adherence to TDF/FTC during OBSP time on study, will be used to interpret the analysis. If substantial differences in HIV incidence are observed between MSM and TGW, consideration will be given to stratifying the Cox regression model by gender identification.

#### 7.3.5 Per-protocol Analysis of Primary Outcome

A per-protocol analysis, excluding participants with exclusionary protocol violations, will be conducted if the number of participants affected exceeds 2% of the enrolled population.

Population: Per Protocol

This analysis will be identical to the mITT analysis specified in section 7.3.3

## 7.3.6 All Follow-Up, Primary Outcome

An analysis of all participants in the mITT cohort, including all follow-up data through the end of the study.

#### 7.4 Safety Analyses

Objective: To compare the safety of oral CAB/CAB LA vs. oral TDF/FTC


#### 7.4.1 Adverse Events

Adverse events: Primary Population: Primary Safety

Descriptive: AEs will be summarized using MedDRA System Organ Class and preferred terms. Tables will show by treatment arm the number and percentage of participants experiencing an AE within a System Organ Class and within preferred term category by severity (grade). For the calculations in these tables, a participant with multiple AEs within a category will be counted once under the maximum severity. Adverse events reported with an onset date prior to the start of treatment will not be considered in the safety analyses. The time windows for consideration of adverse events with onset dates after the discontinuation of treatment are described below (adverse events on Step 1 and Step 2). All adverse events with onset dates within these constraints are considered to be treatment emergent adverse events.

Statistical analysis: Formal statistical comparison of number of safety events across arms is not planned for all events since interpretation of differences must rely heavily upon clinical judgment. Where formal statistical testing is considered necessary to guide judgement of observed differences for any single event or collection of events, differences in events Grade 2 and higher will be assessed. The event rate and 95% confidence interval for each treatment arm will be calculated based on an exact Poisson model, and event rates will be compared between treatment arms using an exact Poisson test.

# Adverse events on blinded study drug product

Objective: To compare the safety of oral CAB/CAB LA vs. oral TDF/FTC while on blinded study drug

Population: Primary Safety

Censoring: For participants who never receive an injection, AEs are censored at the earliest of 1 day after the date of termination or investigational product discontinuation or 120 days after randomization. For participants who receive an injection, AEs are censored at earliest of: open label TDF/FTC first dispensed, 6 weeks after injection if only one injection is given or 10 weeks after the last injection received if 2 or more injections are given. If a termination or product discontinuation occurs, Reported AEs will be excluded if they occur after the censoring time. Details of the OBSP safety censoring definitions are given in Appendix C.

Descriptive and statistical analyses will be as described for Primary Safety above.

## Adverse events in Step 1

Objective: To compare the safety of oral CAB vs. oral TDF/FTC in Step 1

Population: Primary Safety

Censoring: For participants who never received an injection AEs are censored at the first of 1 day after the date of termination or investigational product discontinuation or 120 days after randomization. For participants who receive an injection, AEs are censored at date of first injection. Reported AEs will be excluded if they occur after the censoring time.


Descriptive and statistical analyses will be as described for Primary Safety above.

Adverse events Step 2 only

Objective: To compare the safety of CAB LA vs. oral TDF/FTC while on blinded injectable study drug

Population: Step 2 safety

Censoring: AEs are censored at 6 weeks after the first infection if only one injection is given, or 10 weeks after the time of the last blinded injection if 2 or more injections are given. Details of the OBSP Safety censoring definitions are given in Appendix C. Reported AEs will be excluded if they occur before the first injection or after the OBSP Safety censoring time.

Descriptive and Statistical Analysis will be performed as described for Primary safety above.

#### 7.4.2 Laboratory evaluations

Population: Primary Safety

Descriptive: Laboratory findings for CBC, chemistries (urea, creatinine, CPK, glucose, calcium, phosphorous, amylase, lipase), liver function (AST, ALT, total bilirubin, alkaline phosphatase) and fasting lipid profile (total cholesterol, triglycerides, HDL, LDL) will be reported by grade, as defined in the "Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events". The proportion of laboratory findings qualifying as Grade 2 or above will be presented. Laboratory values will be reported by arm as median, 1st and 3rd quartiles, min and max, and (at follow-up visits) as median, 1st and 3rd quartile change from baseline (see below). Summaries involving values and changes from baseline at scheduled visit time points will consider values from scheduled visits only, and in the case of missing values, results will not be carried forward from interim (unscheduled) visits. For summaries and analyses involving changes in laboratory values over time or maximum change from baseline (e.g. shift tables), values from interim (unscheduled) visits will also be considered.

Formal comparisons of laboratory values will be conducted as follows:

- 1) Absolute values: A mixed-effects model with participant as the random effect and site and arm as fixed effects will be used to assess overall differences in each laboratory outcome by arm. A continuous time (elapsed study time) term and an interaction term with study arm will be added to model time trends in laboratory values that may emerge with continuous exposure to study drug. Only post baseline visits will be included.
- 2) Change from baseline. A fixed effect model with site and arm as covariates will be used to assess overall in change from baseline value for each laboratory outcome by arm. A continuous time (elapsed study time) term interaction with study arm will be added to model differences in laboratory values that may emerge with continuous exposure to study drug.

# Laboratory evaluations while on blinded study drug

Population: Primary Safety

Censoring: Lab assessments are censored at 120 days after enrollment for participant who never receive an injection; at open label FTC/TDF first dispensed, or 10 weeks after


the last injection (6 weeks if only one injection is given), whichever occurs first, otherwise. Laboratory evaluations will be excluded if they occur after the censoring time.

Descriptive and Statistical Analysis as described for Laboratory Evaluations above.

# 7.4.3 Time to study-product discontinuation

Population: mITT

Descriptive: The number and proportion of study participants who discontinue study product will be tabulated by time on study. A Kaplan Meier-type plot of time to first discontinuation will depict the proportion of participants with product discontinuation after randomization, by arm. Competing risk methods will be used to describe the proportion of discontinuation occurring due to safety concern, participant refusal, loss to follow-up or other reasons.

#### Analysis:

Discontinuation for safety: For the purposes of this analysis, study-product discontinuation for safety is defined as a clinical discontinuation prescribed by site clinicians, site staff, or the study CMC for reasons related to participant safety. For study participants who discontinue study medication on their own, or who are discontinued for reasons other than safety, discontinuation events will be treated as competing risks. A competing-risks model (6), stratified by region with study arm as the only covariate will be used to estimate the relative risk comparing the risk of safety discontinuation in Arm A (oral CAB/CAB LA) to Arm B (oral TDF/FTC) and generate the 95% Wald-based confidence interval. Non-safety related discontinuations will be treated as competing-risk events.

Discontinuation for any reason: For the purposes of this analysis, discontinuation of blinded study product for any reason, including loss to follow-up, will be included as an event. A Cox proportional hazard model, stratified by region with study arm as the only covariate will be used to estimate the relative risk comparing the risk of study product discontinuation in Arm A (oral CAB/CAB LA) to Arm B (oral TDF/FTC) and generate the 95% Wald-based confidence interval.

Details of definitions for safety and other reasons are given in Appendix D.

#### 7.5 Secondary Analyses

# 7.5.1 Objective: To compare HIV incidence among participants randomized to CAB LA injections vs. oral TDF/FTC in Step 2 only

Population: STEP 2 Efficacy

Descriptive analyses: These parallel the descriptive analyses described in 7.3.3.

Statistical Analysis: This analysis exactly parallels the Primary ITT analysis, but includes only participants who receive an injection, with Time 0 starting at the time of the first injection (first active injection for the CAB LA arm or first placebo injection for the TDF/FTC arm). The statistical hypothesis being tested for Step 2 remains the same as the primary analysis. A sensitivity analysis using on blinded study product censoring time will follow the same plan as the primary analyses.

# 7.5.2 Objective: To compare HIV incidence among participants randomized to CAB LA injections vs. oral TDF/FTC (Steps 1, 2, and 3 combined)

Population: mITT


Descriptive analyses: These parallel the descriptive analyses in 7.3.3.

Censoring time: First of HIV seroconversion date or last HIV test conducted on study.

Statistical Analysis: This analysis will exactly parallel the Primary ITT analysis, but include all available study follow-up. No formal hypothesis test is proposed for this analysis, as similar infection rates are expected between both arms during Step 3 which could decrease incidence-rate differences between treatment arms.

# 7.5.3 Objective: To compare HIV incidence among participants randomized to CAB LA injections vs. oral TDF/FTC while taking open label TDF/FTC (Step 3 only, descriptive)

Population: STEP 3 Efficacy

Descriptive analyses: These parallel the descriptive analyses in 7.3.3

Statistical Analysis: This analysis will parallel the Primary analysis, but restricted to the study follow-up in after Week 153 (Step 3), with Time 0 set to the beginning of Step 3. Similar infection rates are expected between both arms during Step 3, although because of limited follow-up time the analysis is not powered to establish equivalence.

# 7.5.4 Objective: To compare the change in risk of HIV acquisition between CAB and oral TDF/FTC strategies (Arm A and Arm B) as participants progress from Step 2 to Step 3

Population: mITT

Analysis: Analysis of this objective will be descriptive, based on HIV incidence rates observed by study step. Study-arm specific incidence rates will be computed separately for Step 2 and Step 3, along with 95% confidence intervals. Definitions of Step 2 and Step 3 study time will follow the definitions used in the STEP2 and STEP 3 population.

# 7.5.5 Objective: To compare HIV incidence among the subgroups of participants randomized to oral CAB/CAB LA vs. oral TDF/FTC by region, age, race, ethnicity, baseline risk, and gender identity

Population: mITT

Subgroup Definitions:

Region: USA/Latin America/Asia and Africa

Age: <30/≥30 years old

Race/Ethnicity: Black/Hispanic/White/Other

Baseline risk:

</> median number of sexual partners

</> median report of condomless receptive anal sex

Gender identity: MSM/TGW

Descriptive analyses: These parallel the descriptive analyses described in Section7.3.3, presented for each of the subgroups defined above.

Analysis: The analysis will parallel the primary analysis, with hazard ratios estimated and reported within each subgroup defined by these baseline covariates. Formal tests of subgroup-by-arm interaction will be used to assess for the presence of effect


modification. On blinded study product analyses, if conducted, will parallel those described for the primary outcome analysis.

# 7.5.6 Objective: To compare changes in renal function, liver function, and bone mineral density (BMD) among participants receiving oral CAB/CAB LA vs. oral TDF/FTC

Population: Primary Safety

Endpoints:

- Serum creatinine
- Creatinine clearance (estimated GFR by Cockcroft gault equation)
- ALT
- AST
- Alk Phosphate
- Total bilirubin
- Bone Mineral Density parameters Z-score at hip and spine

Descriptive analysis: As previously described in Section 7.4.2, Laboratory values will be reported by arm as median, 1<sup>st</sup> and 3<sup>rd</sup> quartiles, min and max, and (at scheduled follow-up visits) median, 1<sup>st</sup> and 3<sup>rd</sup> quartile change from baseline.

Statistical Analysis: Each outcome measure will be assessed in two separate models. For each outcome variable all non-missing values will be modeled using mixed-effects regression for correlated data with participant as a random effect. In Model 1 the outcome measure will be change from baseline, and the model will include fixed effects for site and treatment arm; a treatment arm by study time interaction will be used. In Model 2 the outcome measure will be absolute levels of the lab measurement (vs change from baseline) and the model will include fixed effects for site, treatment arm, time (continuous, days from enrollment), and treatment arm by time interaction. Model 2 will assess any difference in time trend between the treatment arms. Log transformations will be used for lab values that show strongly skewed distributions. Nonlinear terms for time will be considered if the time trends appear to be non-linear.

# 7.5.7 Objective: To evaluate and compare rates of HIV drug resistance among participants who acquire HIV infection during the study among participants receiving oral CAB/CAB LA vs oral TDF/FTC

Population: SEROCONVERTERS

Descriptive analysis: The number of participants with HIV drug resistance at the first HIV positive visit will be identified by the presence of mutations known to be associated with CAB (including T66I, E92Q/M, F121Y, Y143R/H/C, S147G, Q148H/K/R, N155H, T97I/A, G140S, and a 5AA duplication at 232), and associated with TDF/FTC (including K65R, K70E, M184V/I) and non-study drugs (all others). Samples from subsequent study visits may also be analyzed, and summaries of resistance and drug concentrations at the visit will be reported. Resistance will be reported separately for those infected prior to enrollment, and during primary analysis follow-up, compared to Step 3.


Statistical Analysis: Proportion of seroconverter participants who have drug-resistance mutations associated with CAB or TDF/FTC at the first HIV positive visit, will be compared between study arms using chi-squared tests (or exact binomial tests when sample size is small). Similar data from subsequent study visits may also be analyzed.

# 7.5.8 Objective: To compare the acceptability of and preferences for CAB LA vs. oral TDF/FTC

Population: mITT

Outcomes:

Primary preference outcome: Responses to whether participants prefer injections over oral tablets (Yes/No)

Primary acceptability outcome: Responses to whether participants feel that the injections/oral tablets are satisfactory (6 point Likert scale).

An additional set of questions are asked about the reasons for medication preference. An additional 12 satisfaction questions are asked for each medication (6 point Likert scale).

Descriptive analysis: Responses to each preference and satisfaction question overall and at each time period will be tabulated and compared across assigned treatment groups.

#### Statistical Analysis:

Chi-square tests and Fisher-exact tests will be used as appropriate, with Likert-scale date converted to binary variables according to distributions within the observed response levels (e.g. at the median response). Time trends will also be evaluated. Inference for differences by arm and trends in time will be analyzed using logistic regression models with GEE estimation to account for intra-participant correlation. Each model will contain four terms: (1) region, (2) time, (3) randomized study arm, and (4) time by arm interaction. Time will be entered into the model as a continuous variable scaled in years. A secondary analysis will evaluate non-linear time trends by entering the time variable into the model as a categorical factor.

# 7.5.9 Objective: To compare changes in weight, blood pressure, pulse, fasting glucose, and fasting lipids among participants receiving oral CAB/CAB LA vs. oral TDF/FTC

Population: Primary Safety

Outcomes:

- Weight,
- BMI
- Blood pressure,
- Pulse,
- Fasting glucose,
- Fasting lipids

Statistical Analysis:


Change from baseline (enrollment) for each outcome will be computed at each follow-up visit where these measures are collected. The mean changes will be plotted over time by treatment arm. A linear mixed model will be fit with categorical intervals for time in study, treatment and time by treatment interaction to evaluate time trends in each arm and the association between treatment and biological measures. Categorical models will also be used to assess changes over time in BMI category, proportion of participants with 5% or more weight change, and occurrence of new diabetes diagnoses. Differences in time trends and treatment effects will be explored for demographic and clinical subgroups, including race/ethnicity, age, baseline smoking status, baseline BMI, and baseline weight.

#### 8. MISSING DATA AND IMPUTATIONS

Data may be missing due to participant dropout, participant nonresponse, missed visits or failures in data collection. In general, the last category (failures in data collection) is quite rare in HPTN trials. Further, it is common to assume that such data are missing completely at random (MCAR) (7) and so will not bias results. However, participant dropout and/or nonresponse are unlikely to be MCAR and so attention must be paid to the potential for bias if there are high levels of missing data for these reasons. Here we discuss the approaches we will take for analyses in the presence of missing data.

For the primary endpoints, HIV infections, safety events, and other biological endpoints, the primary cause of missing data is missed visits and participant dropout. Historically, HPTN trials have had good retention of participants and we expect that to be the case for this trial. Therefore, analyses will be conducted assuming uninformative censoring. If loss-to-follow-up is low and similar between the arms we will not conduct any additional sensitivity analyses. However, if loss-to-follow-up is greater than 20% or meaningfully different between arms (>5%-points), then we will investigate the sensitivity of the results to assumptions about the missing data. Specifically, we will use inverse probability-of-censoring weights to adjust for loss-to-follow-up (8) and compare the adjusted treatment effect to the unadjusted treatment effect. In addition, we will perform a tipping-point analysis whereby we will determine the difference from the observed treatment arm effect (either higher or lower than observed) that would have to exist in the missing data to meaningfully change our interpretation of the results. We will also estimate the difference in treatment-arm effect that would be observed if all participants who are lost-to-follow-up are assumed to have stopped taking PrEP.

Behavioral and self-reported endpoints (e.g. acceptability) may also be subject to participant nonresponse. The analyses described below are based on a complete case approach. However, if non-response is high (>15%) or differential between arms (> 5%-points) then we will perform sensitivity analyses using multiple imputation. Baseline data will be used to develop the imputation model and standard errors will be adjusted using Rubin's method (9). Both complete case and multiple imputation results will be reported.

# 8.1 Missing Start and Stop Dates for Prior and Concomitant Medication, and Medical History

Start date:

- 1. If start date is completely missing, start date will not be imputed.
- 2. If (year is present and month and day are missing) or (year and day are present and month is missing), set month and day to January 1.
- 3. If year and month are present and day is missing, set day to the 1st day of month.


# Stop date:

- 1. If end date is completely missing, end date will not be imputed.
- 2. If (year is present and month and day are missing) or (year and day are present and month is missing), set month and day to December 31st.
- 3. If year and month are present and day is missing, set day to the last day of month.

# 8.2 Missing Start and Stop Dates for Adverse Events

#### Start date:

- 1. If start date is completely missing, start date is set to date of first dose.
- 2. If (year is present, and month and day are missing) or (year and day are present and month is missing):
  - a. If year = year of first dose, then set month and day to month and day of first dose.
  - b. If year < year of first dose, then set month and day to December 31st.
  - c. If year > year of first dose, then set month and day to January 1st.
- 3. If month and year are present and day is missing:
  - a. If year = year of first dose and
    - i. If month = month of first dose, then set day to day of first dose date.
    - ii. If month < month of first dose, then set day to last day of month.
    - iii. If month > month of first dose, then set day to 1st day of month.
  - b. If year < year of first dose, then set day to last day of month.
  - c. If year > year of first dose, then set day to 1st day of month.

#### Stop date:

If the outcome of the AE was ongoing or unknown, then the rules outlined below will not be applied.

- 1. If stop date is completely missing, stop date is set to date of study discontinuation.
- 2. If (year is present, and month and day are missing) or (year and day are present, and month is missing):
  - a. If year = year of study discontinuation, then set month and day to month and day of study discontinuation.
  - b. If year < year of study discontinuation, then set month and day to December 31st.
  - c. If year > year of study discontinuation, then set month and day to December 31st.
  - d. If date created from imputation is after study discontinuation, date of discontinuation will be used
- 3. If month and year are present and day is missing:
  - a. If year = year of study discontinuation and
  - b. If month = month of study discontinuation, then set day to day of study discontinuation date.
    - i. If month < month of study discontinuation, then set day to last day of month
    - ii. If month > month of study discontinuation, then set day to last day of month.
    - iii. If year < year of study discontinuation, then set day to last day of month.
  - c. If year > year of study discontinuation, then set day to last day of month.


#### 9. MONITORING REPORTS

#### 9.1 Performance Metric Reports

Real-time performance metric reports will be available to the protocol team. The content of these reports will be developed by the protocol team and will generally include the following information, overall and by site:

Open Reports for the protocol team

- 1. Accrual
- 2. Demographics
- 3. Rates of progression from Step 1 to Step 2
- 4. Retention
- 5. Rates of continuation on study medications
- 6. Data completeness and timeliness

#### 9.2 SMC Reports

Monitoring reports will be provided to the HPTN Study Monitoring Committee (SMC) approximately every six months (see HPTN SMC Charter). The content of these reports will be developed by the protocol team, but will generally include the following information, overall and by site:

#### Open Report

- 1. Screening
- 2. Accrual
- 3. Baseline demographic characteristics of enrolled participants
- 4. Baseline self-reported HIV risk behavior
- 5. Disposition
- 6. Retention (Step 1, Step 2, Step 3 separately)
- 7. Adherence to injection regimen, receipt of oral pills
- 8. Lost-to-follow-up, Withdrawal, Termination, Product Holds, Death (excluding those attributed to potential HIV infection)
- 9. Protocol deviations
- 10. DMQ and Lab Center report

# Closed Report

1. HIV incidence rate by region, aggregated over study arm.

#### 9.3 DSMB Reports

Monitoring reports will be provided to the DSMB approximately every six months or as requested by the DSMB. DSMB review will occur at a minimum once per year. At any DSMB meeting, or at any time between regularly scheduled meetings, the DSMB may alter the reporting schedule and request an additional meeting and/or report or request a


change to the meeting schedule. The contents of the DSMB reports will be detailed elsewhere (see DSMB Report Table of Contents), but will generally include the following:

## Open Report:

1. All tables and figures in the SMC report.

#### Medical Officer Report

- 1. Grade 3 and above adverse events, aggregated by arm
- 2. SAEs, aggregated by arm
- 3. Injection Site Reactions, aggregated by arm

#### Closed report

- 1. Interim TDF/FTC adherence monitoring results
- 2. Adverse events and Injection Site Reactions, by arm
- 3. Summary of the primary outcome data (HIV incidence) by arm
- 4. At formal interim monitoring review, Interim Endpoint Analysis of the primary ITT outcomes, including pre-planned group-sequential stopping boundaries.
- 5. OBSP analyses of the primary outcomes
- 6. Descriptive tables of the timing of infections relative to injections for HIV infections in the CAB arm.

## 9.4 Clinical Study Report

The tables described below will be included in the CSR. Additional tables and analyses may be included, at the discretion of the protocol team or sponsor, e.g., depending on the availability of additional laboratory evaluations. All reports and analyses will be presented by study arm.

- 1. Participant Disposition
- 2. Screening Status
- 3. Study Populations Summary
- 4. Subject Status and Accountability
- 5. Protocol Deviations
- 6. Demographic and Baseline Variables
- 7. Concurrent Illnesses and Medical Conditions
- 8. Prior and Concurrent Medications
- 9. Adherence to Blinded Study Medication
- 10. Exposure to Blinded Study Medication and Needle Size Summaries
- 11. Sexually Transmitted Infection Summaries
- 12. Safety

Adverse events (including injection site reactions) will be summarized in the following reports:


- Overall Summaries of AEs
- Incidences of AEs
- Severity of AEs
- o Relationship of the AEs to the Randomized Treatment
- Serious Adverse Events
- Adverse Events Leading to Drug Withdrawal
- Adverse Events with Study Steps
- Overall Summary of Adverse Events of Special Interest

*Note*: Adverse Events of Special Interest will be detailed separately in an Integrated Summary of Safety (ISS)

- 13. Safety Laboratory Data: Summaries and shift tables: Hematology, Renal Function, Liver Function, Lipid Profiles, Urinalysis, Other Clinical Chemistry, Laboratories Meeting Stopping Criteria
- 14. Vital Signs, including weight, BMI, BP, pulse, fasting glucose/lipids

Note: Descriptive statistics only; no formal statistical comparisons included in the CSR

- 15. Efficacy Analyses and Summaries
- 16. Self-Reported Risk Behaviors

Note: Descriptive statistics only; no formal statistical comparisons included in the CSR

17. Satisfaction, Attitudes, and Preferences Assessments

Note: Descriptive statistics only; no formal statistical comparisons included in the CSR

18. FTC/TDF PK assessments of the adherence cohort (Plasma, DBS)

*Note*: Descriptive statistics only; no formal statistical comparisons included in the CSR Cabotegravir PK assessments in a subpopulation

Note: Descriptive statistics only; no formal statistical comparisons included in the CSR

19. PK assessments of seroconverters

Note: Descriptive statistics only; no formal statistical comparisons included in the CSR

20. Resistance assessment of seroconverters

Note: Descriptive statistics only; no formal statistical comparisons included in the CSR

21. Planned/Unplanned Participant Unblinding Events

#### 10. Revisions of the SAP

# 10.1. Changes in version 2.0 of the SAP

# Revisions prompted by changes in Version 2.0 and 3.0 of the protocol

- Change from open ended follow-up to maximum follow-up of 3 years per person.
- Increase of sample size from 4500 to 5000 participants


#### Revisions prompted by results external to the protocol

- Addition of new objective: To compare changes in weight, blood pressure, pulse, fasting glucose and fasting lipids among participants receiving oral CAB/CAB LA vs. oral TDF/FTC
- Removal of the upper limit of 1.23 for the non-inferiority margin in the sensitivity analysis adapted to the FTC/TDF adherence observed in the study cohort.
- Two separate As treated analyses replaced by a single On Blinded Study Product analysis. This reduces and simplifies the number of sensitivity analyses proposed for the study.
- Change in emphasis of analysis recomputing the NI margin from sensitivity analysis to a supportive analysis.

### Revisions related to alignment with the SAP template adopted by SCHARP

- Added signature page
- Addition of Sections on sample size and power, randomization, blinding
- Addition of pre-defined subgroups
- General rearrangement of sections and renumbering.
- Addition of section describing treatment of missing data

# Revisions related to study data collection and/or conduct

- On study drug definition changed to align with injection delivery for both arms. Data
  about availability of pills in participants assigned to the FTC/TDF arms is too
  incomplete to accurately characterize potential adherence. In addition, the use of the
  same metric in both arms will likely reduce ascertainment bias.
- Removal of ongoing assessment of CAB concentration within seroconverters, to reduce the risk of inadvertent release of information about relative efficacy.
- Change study time contributed for seroconverters from time HIV infection detected to midpoint of interval in which seroconversion detected. This is to lessen the impact of different study schedules.

# Revisions related to sponsor/DSMB requests

- Clarification of the information reported in Open, Medical Officer and Closed reports
- Clarification of the information reviewed by the HPTN SMC

#### 10.2 Changes in version 3.0 of the SAP

Version 3.0 was prepared following the decision to unblind the study results following the May 14 2020 review. The unblinded statistician continued to not have access to individual level data.

#### **Revisions to Safety**

The safety population was revised to include safety observed in the oral lead-in (Section 6.6), and definitions of Step 1 and Step 2 safety populations.


#### Revision to interim monitoring

Interim monitoring guidance to stop for efficacy revised to stop for evidence of non-inferiority, i.e. monitoring against the trial null hypothesis H0: HR (CAB vs FTC/TDF) > 1.23. (Section 7.2.2)

# Reorganization of sections and new sections

- Added Abbreviation and Definition Section
- Reorganized existing text into a new Section 4 Statistical Considerations which includes Randomization, Blinding & Sample Size and Power for the Study.
- Changed the Name of Section 4 (now section 5) Blinded Review of HIV and Protocol Exclusion to Blinded Review of HIV and Protocol Violations
- Changed the name of Section 5 (now section 6) from General Data Analysis Considerations to Analysis Population.
  - o Added definition of STEP 1 population
- Reorganized existing text into a new Section 7 Statistical Analyses which includes Interim Analyses (previously Section 5), Efficacy Analyses (previously Section 8), Safety Analyses (previously Section 9) and Secondary Analyses (previously Section 10)
- Added a new Section 8 Missing Data and Imputation
- In Section 9 Monitoring Reports Added description of Clinical Study Report.

# 10.3 Changes in version 4.0 of the SAP

Version 4.0 was prepared during the planning process for the Clinical Study Report. The unblinded statistician continued to have no access to individual level data.

#### **Analysis Populations**

- Populations were renamed or clarified: ITT renamed mITT; Step 1 and 2 Safety, Step 2 Efficacy, Seroconverter populations.
- Populations were added: ITT; Longitudinal Pharmacology for cabotegravir.
- Populations were deleted: Step 1 Efficacy, All Follow-up.
- Populations were respecified as censoring schemes: On blinded study product.

# **Analysis Details and Clarifications**

- Clarifications and additional details were added throughout the Statistical Analysis section. These included:
  - o definitions of AE onset windows and censoring times added to safety analyses;
  - details added regarding analyses of change from baseline laboratory values;
  - o references to "South America" changed to "Latin America";
  - clarification to stop-date imputation algorithm;
- Appendices were added to provide detail for visit windowing, key subpopulations, efficacy analysis details, censoring and OBSP specifications, study drug discontinuation analysis, and a listing of adverse events of special interest (AESI).


#### Reports

Updates were made to the Clinical Study Report contents

# **CHANGE HISTORY**

| Version | | Affected | Activity Description |
|---|---|---|---|
| Number | Effective Date | Section(s) | 3 |
| 2.0 | April 17, 2020 | All Sections | Update to ensure sections are in compliance with SCHARP SAP template. Substantive reviews as a result of changes detailed in Section 10.1. |
| 3.0 | July 01, 2020 | Sections<br>5.1.2 and 6.2 | Updated to reflect the change to interim monitoring based on non-inferiority margins (in revised Interim Monitoring Guidance v 2.0 (08May2020). Updated to included oral lead-in in safety population. Minor updates and reorganization as detailed in Section 15.7. |
| 4.0 | October 02,<br>2020 | Throughout<br>Sections 6<br>and 7; 9.3;<br>Appendices | Clarifications and updates to Analysis Populations and subgroups. Additional details in definitions of censoring. Other updates as detailed in Section 10.3 |

#### References

- 1. McCormack S, Dunn DT, Desai M, Dolling DI, Gafos M, Gilson R, et al. Pre-exposure prophylaxis to prevent the acquisition of HIV-1 infection (PROUD): effectiveness results from the pilot phase of a pragmatic open-label randomised trial. Lancet. 2016;387(10013):53-60.
- 2. Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, et al. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. The New England journal of medicine. 2010;363(27):2587-99.
- 3. Molina JM, Charreau I, Chidiac C, Pialoux G, Cua E, Delaugerre C, et al. Post-exposure prophylaxis with doxycycline to prevent sexually transmitted infections in men who have sex with men: an open-label randomised substudy of the ANRS IPERGAY trial. Lancet Infect Dis. 2018;18(3):308-17.
- 4. Draft FDA Guidance Document. Guidance for industry non-inferiority clinical trials. In: FOOD AND DRUG ADMINISTRATION DOHAHS, editor. 2010.
- 5. Hanscom B, Hughes JP, Williamson BD, Donnell D. Adaptive non-inferiority margins under observable non-constancy. Stat Methods Med Res. 2018:962280218801134.
- 6. Fine JP, Gray RJ. A Proportional Hazards Model for the Subdistribution of a Competing Risk. Journal of the American Statistical Association. 1999;94(446):496-509.
- 7. Little RJA, Rubin DB. Statistical analysis with missing data. 2nd ed. Hoboken, N.J.: Wiley; 2002. xv, 381 pages p.
- 8. Cain LE, Cole SR. Inverse probability-of-censoring weights for the correction of time-varying noncompliance in the effect of randomized highly active antiretroviral therapy on incident AIDS or death. Stat Med. 2009;28(12):1725-38.
- 9. Rubin DB. Multiple imputation for nonresponse in surveys. New York: Wiley; 1987. xxix, 258 pages p.


Protocol HPTN 083 Statistical Analysis Plan

# **Appendix A Visit windows**HPTN 083 Visit Codes, Target Days, and Visit Windows

| Week | Visit Code | Target day | Target visit<br>window<br>(±varies days) | Allowable visit<br>window<br>(± varies days) | Allowable visit window |
|---|---|---|---|---|---|
| Screening | 1.0 | | | , | |
| | | S | tep 1 | | |
| Day 0/Enrollment | 2.0 | 0 | (0,3) | +6 | (0,6) |
| Week 2 | 3.0 | 14 | (11, 17) | -7 / +6 | (7, 20) |
| Week 4 | 4.0 | 28 | (25, 31) | -7 / +3 | (21, 31) |
| | | S | tep 2 | | , , , |
| Week 5 | 5.0 | 35 | (32, 38) | -3 / +3 | (32 . 38) |
| Week 6 | 6.0 | 42 | (39, 45) | -3 / +10 | (39, 52) |
| Week 9 | 7.0 | 63 | (60 . 66) | -10 / +3 | (53 . 66) |
| Week 10 | 8.0 | 70 | (67, 73) | -3 / +24 | (67, 94) |
| Week 17 | 9.0 | 119 | (112 , 126) | -24 / +7 | (95 , 126) |
| Week 19 | 10.0 | 133 | (127 , 140) | -6 / +20 | (127,153) |
| Week 25 | 11.0 | 175 | (168 , 182) | -21 / +7 | (154 ,182) |
| Week 27 | 12.0 | 189 | (183, 196) | -6 / +20 | (183, 209) |
| Week 33 | 13.0 | 231 | (224, 238) | -21 / +7 | (210, 238) |
| Week 35 | 14.0 | 245 | (239, 252) | -6 / +20 | (239, 265) |
| Week 41 | 15.0 | 287 | (280, 294) | -21 / +7 | (266, 294) |
| Week 43 | 16.0 | 301 | (295, 308) | -6 / +20 | (295, 321) |
| Week 49 | 17.0 | 343 | (336, 350) | -21 / +7 | (322, 350) |
| Week 51 | 18.0 | 357 | (351, 364) | -6 / +20 | (351, 377) |
| Week 57 | 19.0 | 399 | (392, 406) | -21 / +7 | (378, 406) |
| Week 59 | 20.0 | 413 | (407, 420) | -6 / +20 | (407, 433) |
| Week 65 | 21.0 | 455 | (448, 462) | -21 / +7 | (434, 462) |
| Week 67 | 22.0 | 469 | (463, 476) | -6 / +20 | (463, 489) |
| Week 73 | 23.0 | 511 | (504, 518) | -21 / +7 | (490, 518) |
| Week 75 | 24.0 | 525 | (519, 532) | -6 / +20 | (519, 545) |
| Week 81<br>Week 83 | 25.0<br>26.0 | 567<br>581 | (560 , 574)<br>(575 , 588) | -21 / +7<br>-6 / +20 | (546 , 574) |
| | | | | | (575, 601) |
| Week 89<br>Week 91 | 27.0<br>28.0 | 623<br>637 | (616, 630)<br>(631, 644) | -21 / +7<br>-6 / +20 | (602, 630)<br>(631, 657) |
| Week 97 | 29.0 | 679 | (672, 686) | -21 / +7 | (658, 686) |
| Week 99 | 30.0 | 693 | (687, 700) | -6 / +20 | (687, 713) |
| Week 105 | 31.0 | 735 | (728 , 742) | -21 / +7 | (714, 742) |
| Week 107 | 32.0 | 749 | (743, 756) | -6 / +20 | (743, 769) |
| Week 113 | 33.0 | 791 | (784, 798) | -21 / +7 | (770, 798) |
| Week 115 | 34.0 | 805 | (799, 812) | -6 / +20 | (799, 825) |
| Week 121 | 35.0 | 847 | (840 , 854) | -21 / +7 | (826 , 854) |
| Week 123 | 36.0 | 861 | (855, 868) | -6 / +20 | (855 , 881) |
| Week 129 | 37.0 | 903 | (896, 910) | -21 / +7 | (882, 910) |
| Week 131 | 38.0 | 917 | (911, 924) | -6 / +20 | (911, 937) |
| Week 137 | 39.0 | 959 | (952, 966) | -21 / +7 | (938, 966) |
| Week 139 | 40.0 | 973 | (967, 980) | -6 / +20 | (967, 993) |
| Week 145 | 41.0 | 1015 | (1008, 1022) | -21 / +7 | (994, 1022) |
| Week 147 | 42.0 | 1029 | (1023, 1036) | -6 / +20 | (1023, 1049) |
| Week 153 | 43.0 | 1071 | (1064, 1078) | -21 / +7 | (1050 , 1078) |
| Week 155 | 44.0 | 1085 | (1079 , 1092) | -6 / +20 | (1079 , 1105) |
| Week 161 | 45.0 | 1127 | (1120 , 1134) | -21 / +7 | (1106 , 1134) |
| Week 163 | 46.0 | 1141 | (1135 , 1148) | -6 / +20 | (1135 , 1161) |
| Week 169 | 47.0 | 1183 | (1176 , 1190) | -21 / +7 | (1162 , 1190) |
| Week 171 | 48.0 | 1197 | (1191 , 1204) | -6 / +20 | (1191 , 1217) |
| Week 177 | 49.0 | 1239 | (1232 , 1246) | -21 / +7 | (1218 , 1246) |
| Week 179 | 50.0 | 1253 | (1247 , 1260) | -6 / +20 | (1247 , 1273) |
| Week 185 | 51.0 | 1295<br>1309 | (1288 , 1302) | -21 / +7 | (1274 , 1302) |
| Week 187 | 52.0 | | (1303 , 1316) | -6 / +20 | (1303 , 1329) |
| Step 3 | | | | | |


HPTN 083 Statistical Analysis Plan

| Day 0 (Step 3 only) | 53.0 | <8 weeks from last injection | (0 , 14) | +42 | (0 , 42) |
|---|---|---|---|---|---|
| Week 12 | 54.0 | 84 | 70, 98 | -41 / +42 | (43, 126) |
| Week 24 | 55.0 | 168 | 154, 182 | -41 / +42 | (127, 210) |
| Week 36 | 56.0 | 252 | 238, 266 | -41 / +42 | (211, 294) |
| Week 48 | 57.0 | 336 | 322, 350 | -41 / +42 | (295, 378) |

### **Appendix B** Definition of subgroups

- Region: USA, Latin America, Asia, Africa as defined in Appendix E
- Age: 30 vs ≥30 years old
- · Race/Ethnicity:
  - For US sites only: Black vs not Black.
    - Black is defined as Black or African American (AA) or Mixed Race, including Black/AA, or Other that includes free text including any of these terms. Non-Black is any other designation that is not missing.
  - Hispanic vs. Non-Hispanic Directly from CRF asking whether participant considers him/herself to be Latino/a or of Hispanic origin
- Baseline risk:
  - ≤/> median number of sexual partners
  - ≤/> median report of condomless receptive anal sex
- Gender identity: MSM, TGW, and prefer not to answer.
- TGW includes participants who self-identify at enrollment as female, transgender male, transgender female, gender queer, transvestite, gender variant, gender non-conforming, or gender fluid or Other, where the free text or any other mentioned above. Participants who self-identify as gay, bisexual, homosexual are included in the MSM category.


### **Appendix C** Details of Efficacy Analysis Definitions

### **Population Definition:**

### **Modified ITT**

- Participant is randomized
- Participant is HIV un-infected at randomization (determined by EAC)
- Participant does not have a major enrollment violation TBD by independent adjudication

Note: Only participants with at least one follow-up visit (of any type, including safety and interim visits) with HIV status determined after enrollment will contribute study time to the efficacy analysis.

### Censoring for primary efficacy analysis:

- If the study is stopped early, all data from the enrollment visit through the end of blinded injection visits will be included
- If no study-wide transition to Step 3 occurred, all data from the enrollment visit through 3 years plus one month (153\*7+30=1101 days) will be considered.
- If study wide transition to Step 3 occurred
  - For participants who have been enrolled more than three years (153 weeks) prior to study-wide transition to Step 3, all data from enrollment through 1101 days will be considered
  - For participants who have been enrolled fewer than three years prior to study-wide transition to Step 3 and are on blinded study product, all the data from enrollment visit through the next scheduled injection visit in their Step 2 schedule after the Step 3 transition date plus one month (30 days) will be considered.
  - For participants who have been enrolled fewer than three years prior to studywide transition to Step 3 who are not on blinded study product, all the data from enrollment visit through the Step 3 transition date plus one month (30 days) will be considered.

### Calculation of study time:

- If HIV infected, study time will be calculated as the number of days between enrollment and the mid-point between first visit where HIV infection was detected and the most recent prior visit where HIV infection was not detectable, as determined by the EAC.
- If HIV un-infected, study time will be calculated as the number of days between enrollment and the last visit with HIV status at or before the censoring time.

### **Primary endpoint:**

Only infections that are confirmed by the EAC and detected within the analysis
timeframe at the time of the final primary analysis adjudication (date of first positive visit
as determined by the EAC within the analysis timeframe) will be considered. Infections
that are not confirmed by the EAC or that occur out of the analysis timeframe will not be
included as primary endpoints.

### Censoring for on blinded study product (OBSP) efficacy analysis

Participants will be censored the first time an injection is delayed, defined as follows:


• Last non-delayed injection: The earliest of an injection whose subsequent injection is delayed for the first time (i.e. given >6 weeks after the Week 5 injection or >10 weeks after any other injection) or the last injection before a termination or a permanent product discontinuation

- For participants with a delayed injection, follow-up time will be censored at the last visit
  with HIV status determined up through 6 weeks after the Week 5 injection, if that is the
  last non-delayed injection, or 10 weeks after the last non-delayed injection for
  subsequent injections.
- For participants with no delayed injections, analysis time defined as for primary efficacy analysis

### Censoring for OBSP Safety analyses

For a participant who never receives an injection, AEs will be censored when the onset date falls after the earliest of 120 days after randomization or at the termination or permanent product discontinuation date +1.

For participants who receive an injection, adverse event follow-up will be censored after the last injection regardless of any delays in injections. If only one injection is given, the participants safety events will be censored at 6 weeks after the injection, or 10 weeks after the last injection if more than one injection is given.

### Interim Analysis (mITT and OBSP) specification

Interim analysis procedures will follow the primary analysis definitions above with the exception that the analysis timeframe will be truncated at the interim-analysis data cut date, as follows.

### Interim mITT analysis

- For participants who have been enrolled at least 1101 days at the time of data cut, all data from enrollment through 1101 days will be considered
- For participants who have been enrolled fewer than 1101 days at the time of data cut, all available data from the enrollment visit through the data cut date will be considered.

### Interim OBSP analysis

- If there is an injection delay prior to the data cut, all data up to the last visit with HIV status determined that occurred prior to the data cut date and within 6/10 weeks for the first/subsequent injection of the last non-delayed injection will be considered.
- If there is no injection delay prior to the data cut point, data included as for the ITT analysis


# Appendix D Study drug discontinuation analysis due to safety

### Definition of Censoring used in analysis of discontinuations due to safety

- Discontinuations due to death, investigator decision and HIV-infection are censored.
- Participants who exit the study at a scheduled exit visit or at the end of the study are also censored.
- Loss to follow-up is treated as a competing event in this analysis: Participants remaining on study product (I.e. in Step 1 or 2) are considered lost to follow-up if
  - (1) participant did not move to step 2 within 60 days of enrollment and has not returned;
  - (2) participant did not receive any injection within 180 days since last injection and has not returned.
- Permanent discontinuation and/or termination due to participant refusal are treated as a competing events, and include: participant unwilling or unable to comply study procedures, injection intolerance, other participant request, or refuse further participation.

### The Safety events of interest are:

 Permanent discontinuation due to safety concerns including: clinical/laboratory AE, ISR, CMC recommendation and other clinical reason.


## **Appendix E** Definitions of Regions for Study Sites

| CRS ID | Region | State/Country | Site Name |
|---|---|---|---|
| 31788 | US | Alabama | Alabama CRS |
| 31957 | Latin America | Argentina | Fundaci¢n Hu'sped CRS |
| 31968 | Latin America | Argentina | Hospital JM Ramos Mejia |
| 12101 | Latin America | Brazil - Rio | Instituto de Pesquisa Clinica Evandro Chagas |
| | | | (IPEC) CRS |
| 12201 | Latin America | Brazil - Porto Alegre | Hospital Nossa Senhora da Conceiâ€jao CRS |
| 31517 | Latin America | Brazil - Sao Paulo | University of Sao Paulo CRS |
| 31954 | Latin America | Brazil - Sao Paulo | Centro Referencia e Treinamento DST/AIDS CRS |
| 601 | US | California | UCLA CARE Center CRS |
| 30305 | US | California | Bridge HIV CRS |
| 31607 | US | California | UCLA Vine Street Clinic CRS |
| 31608 | US | California | George Washington University CRS |
| 31967 | US | California | East Bay AIDS Center (EBAC) CRS |
| 31961 | US | Colorado | Children's Hospital Colorado CRS |
| 5802 | US | Georgia | Ponce de Leon Center CRS |
| 31440 | US | Georgia | Hope Clinic of the Emory Vaccine Center CRS |
| 30347 | US | Illinois | UIC Project WISH CRS |
| 31958 | US | Illinois | Adolescent and Young Adult Research at the CORE Center (AYAR at CORE) |
| 31959 | US | Louisiana | New Orleans Adolescent Trials Unit CRS |
| 201 | US | Maryland | Johns Hopkins University CRS |
| 31785 | US | Massachusetts | Fenway Health (FH) CRS |
| 2101 | US | Missouri | Washington University Therapeutics (WT) CRS |
| 31786 | US | New Jersey | New Jersey Medical School Clinical Research<br>Center CRS |
| 7804 | US | New York | Weill Cornell Chelsea CRS |
| 30261 | US | New York | Bronx Prevention Research Center CRS |
| 30276 | US | New York | Harlem Prevention Center CRS |
| 31801 | US | New York | New York Blood Center CRS |
| 3201 | US | North Carolina | Chapel Hill CRS |
| 3203 | US | North Carolina | Greensboro CRS |
| 2301 | US | Ohio | Ohio State University CRS |
| 2401 | US | Ohio | Cincinnati Clinical Research Site |
| 30310 | US | Pennsylvania | Penn Prevention CRS |
| 11301 | Latin America | Peru | Barranco CRS |
| 11302 | Latin America | Peru | San Miguel CRS |
| 30259 | Latin America | Peru | Asociacion Civil Selva Amazonica (ACSA) CRS |
| 31909 | Latin America | Peru | Via Libre CRS |
| 31970 | Latin America | Peru | Centro de Investigaciones Tecnologicas,<br>Biomedicas y Medioambientales (CITBM) CRS |
| 31708 | Africa | South Africa | Groote Schuur HIV CRS |
| 6501 | US | Tennessee | St. Jude Children's Research Hospital CRS |
| 31473 | US | Texas | Houston AIDS Research Team CRS |
| 31458 | Asia | Thailand | CMU HIV Prevention CRS |
| 31681 | Asia | Thailand | Silom Community Clinic CRS |
| 31802 | Asia | Thailand | Thai Red Cross AIDS Research Centre (TRC-ARC) CRS |
| 31969 | Asia | Vietnam | Yen Hoa Health Clinic |


Appendix F: Adverse Events of Special Interest Hepatotoxicity (Hepatic failure, fibrosis and cirrhosis and other liver damagerelated conditions)

| PT | PT Code |
|----------------------------------------------------|----------|
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cardiohepatic syndrome | 10082480 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10071203 |
| Drug-induced liver injury Duodenal varices | 10072268 |
| Gallbladder varices | 10051010 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Gastrooesophageal variceal haemorrhage prophylaxis | 10066597 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Immune-mediated cholangitis | 10083406 |
| Immune-mediated hepatic disorder | 10083521 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |
| Liver injury | 10067125 |
| Liver operation | 10067125 |


| Liver transplant | 10024714 |
|---------------------------------------|----------|
| Lupoid hepatic cirrhosis | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Nonalcoholic fatty liver disease | 10082249 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Sugiura procedure | 10083010 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |

## Hepatotoxicity Continued (Hepatitis, non-infectious)

| PT | PT Code |
|--------------------------------------------|----------|
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |


| Non-alcoholic steatohepatitis | 10053219 |
|-------------------------------|----------|
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |

### Hyperglycaemia

| пурегдіусаенна | |
|-----------------------------------------------------|----------|
| PT | PT Code |
| Acquired lipoatrophic diabetes | 10073667 |
| Blood 1,5-anhydroglucitol decreased | 10065367 |
| Blood glucose increased | 10005557 |
| Diabetes complicating pregnancy | 10012596 |
| Diabetes mellitus | 10012601 |
| Diabetes mellitus inadequate control | 10012607 |
| Diabetes with hyperosmolarity | 10012631 |
| Diabetic arteritis | 10077357 |
| Diabetic coma | 10012650 |
| Diabetic coronary microangiopathy | 10080788 |
| Diabetic hepatopathy | 10071265 |
| Diabetic hyperglycaemic coma | 10012668 |
| Diabetic hyperosmolar coma | 10012669 |
| Diabetic ketoacidosis | 10012671 |
| Diabetic ketoacidotic hyperglycaemic coma | 10012672 |
| Diabetic ketosis | 10012672 |
| Diabetic ketosis Diabetic metabolic decompensation | 10074309 |
| Diabetic metabolic decompensation Diabetic wound | 10081558 |
| Euglycaemic diabetic ketoacidosis | 10081338 |
| | 10080061 |
| Fructosamine increased | |
| Fulminant type 1 diabetes mellitus | 10072628 |
| Gestational diabetes | 10018209 |
| Glucose tolerance impaired | 10018429 |
| Glucose tolerance impaired in pregnancy | 10018430 |
| Glucose urine present | 10018478 |
| Glycated albumin increased | 10082836 |
| Glycosuria | 10018473 |
| Glycosuria during pregnancy | 10018475 |
| Glycosylated haemoglobin abnormal | 10018481 |
| Glycosylated haemoglobin increased | 10018484 |
| Hyperglycaemia | 10020635 |
| Hyperglycaemic hyperosmolar nonketotic syndrome | 10063554 |
| Hyperglycaemic seizure | 10071394 |
| Hyperglycaemic unconsciousness | 10071286 |
| Impaired fasting glucose | 10056997 |
| Insulin resistance | 10022489 |
| Insulin resistant diabetes | 10022491 |
| Insulin-requiring type 2 diabetes mellitus | 10053247 |
| Ketoacidosis | 10023379 |
| Ketonuria | 10023388 |
| Ketosis | 10023391 |
| Ketosis-prone diabetes mellitus | 10023392 |
| Latent autoimmune diabetes in adults | 10066389 |
| Monogenic diabetes | 10075980 |
| Neonatal diabetes mellitus | 10028933 |
| New onset diabetes after transplantation | 10082630 |
| Pancreatogenous diabetes | 10033660 |
| Steroid diabetes | 10081755 |
| Type 1 diabetes mellitus | 10067584 |
| Type 2 diabetes mellitus | 10067585 |
| Type 3 diabetes mellitus | 10072659 |
| Urine ketone body present | 10057597 |


### **Hypersensitivity Reactions**

| PT | PT Code |
|-------------------------------------------------------|----------|
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Pseudolymphoma | 10037127 |
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |
| Circumoral oedema | 10052250 |
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |
| Periorbital swelling | 10056647 |
| Swelling of eyelid | 10042690 |

### Rash

| PT | PT Code |
|-------------------------------------------------------|----------|
| Acute generalised exanthematous pustulosis | 10048799 |
| Bullous haemorrhagic dermatosis | 10083809 |
| Cutaneous vasculitis | 10011686 |
| Dermatitis bullous | 10012441 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Epidermal necrosis | 10059284 |
| Erythema multiforme | 10015218 |
| Erythrodermic atopic dermatitis | 10082985 |
| Exfoliative rash | 10064579 |
| Oculomucocutaneous syndrome | 10030081 |
| SJS-TEN overlap | 10083164 |
| Skin necrosis | 10040893 |
| Stevens-Johnson syndrome | 10042033 |
| Target skin lesion | 10081998 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |
| Nodular rash | 10075807 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash popular | 10037876 |


| Rash rubelliform | 10057984 |
|---------------------|----------|
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |
| Drug eruption | 10013687 |

Suicide/self-injury

| PT | PT Code |
|-------------------------------------------------|----------|
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |
| Suspected suicide | 10082458 |
| Suspected suicide attempt | 10081704 |

Depression (Exclude suicide and self-injury)

| PT | PT Code |
|-----------------------------------------------------------|----------|
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Depression postoperative | 10012390 |
| Depressive symptom | 10054089 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

Bipolar Disorder

| Dipolal Disolate | |
|----------------------|----------|
| PT | PT Code |
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |


Statistical Analysis Plan HPTN 083

| Mania | 10026749 |
|-------|----------|

| PT | PT Code |
|---|---|
| Acute psychosis | 10001022 |
| Alcoholic psychosis | 10001632 |
| Alice in wonderland syndrome | 10001666 |
| Brief psychotic disorder with marked stressors | 10048549 |
| Brief psychotic disorder without marked stressors | 10056395 |
| Brief psychotic disorder, with postpartum onset | 10006362 |
| Charles Bonnet syndrome | 10063354 |
| Childhood psychosis | 10061040 |
| Clang associations | 10009232 |
| Cotard's syndrome | 10059591 |
| Delusion | 10012239 |
| Delusion of grandeur | 10012241 |
| Delusion of parasitosis | 10012242 |
| Delusion of reference | 10012244 |
| Delusion of replacement | 10012245 |
| Delusion of theft | 10084030 |
| Delusional disorder, erotomanic type | 10012249 |
| Delusional disorder, grandiose type | 10012250 |
| Delusional disorder, jealous type | 10012251 |
| Delusional disorder, mixed type | 10012252 |
| Delusional disorder, persecutory type | 10053195 |
| Delusional disorder, somatic type | 10012254 |
| Delusional disorder, unspecified type | 10012255 |
| Delusional perception | 10012258 |
| Dementia of the Alzheimer's type, with delusions | 10012295 |
| Depressive delusion | 10063033 |
| Derailment | 10012411 |
| Epileptic psychosis | 10059232 |
| Erotomanic delusion | 10015134 |
| Flight of ideas | 10016777 |
| Hallucination | 10019063 |
| Hallucination, auditory | 10019070 |
| Hallucination, gustatory | 10019071 |
| Hallucination, olfactory | 10019072 |
| Hallucination, synaesthetic | 10062824 |
| Hallucination, tactile | 10019074 |
| Hallucination, visual | 10019075 |
| Hallucinations, mixed | 10019079 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hysterical psychosis | 10062645 |
| Ideas of reference | 10021212 |
| Illusion | 10021212 |
| Jealous delusion | 10021403 |
| Loose associations | 10024825 |
| Mixed delusion | 10076429 |
| Neologism | 10076429 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Paranoia | 10073293 |
| Paranoid personality disorder | 10033869 |
| Paranoid personality disorder Parkinson's disease psychosis | |
| Paroxysmal perceptual alteration | 10074835 |
| | 10063117 |
| Persecutory delusion | 10034702 |
| Postictal psychosis Post-injection delirium sedation syndrome | 10070669<br>10072851 |


| Posturing | 10036437 |
|-------------------------------------------------------|----------|
| Psychosis postoperative | 10065617 |
| Psychotic behaviour | 10037249 |
| Psychotic disorder | 10061920 |
| Psychotic disorder due to a general medical condition | 10061921 |
| Reactive psychosis | 10053632 |
| Rebound psychosis | 10074833 |
| Schizoaffective disorder | 10039621 |
| Schizoaffective disorder bipolar type | 10068889 |
| Schizoaffective disorder depressive type | 10068890 |
| Schizophrenia | 10039626 |
| Schizophreniform disorder | 10039647 |
| Schizotypal personality disorder | 10039651 |
| Senile psychosis | 10039987 |
| Shared psychotic disorder | 10040535 |
| Somatic delusion | 10041317 |
| Somatic hallucination | 10062684 |
| Substance-induced psychotic disorder | 10072388 |
| Tangentiality | 10043114 |
| Thought blocking | 10043495 |
| Thought broadcasting | 10052214 |
| Thought insertion | 10043496 |
| Thought withdrawal | 10043497 |
| Transient psychosis | 10056326 |
| Waxy flexibility | 10047853 |

### **Mood Disorders**

| PT | PT Code |
|--------------------------------------------------|----------|
| Affect lability | 10054196 |
| Affective ambivalence | 10077173 |
| Affective disorder | 10001443 |
| Alexithymia | 10077719 |
| Anger | 10002368 |
| Apathy | 10002942 |
| Blunted affect | 10005885 |
| Boredom | 10048909 |
| Constricted affect | 10010778 |
| Crying | 10011469 |
| Diencephalic syndrome of infancy | 10012774 |
| Dysphoria | 10013954 |
| Emotional disorder | 10014551 |
| Emotional distress | 10049119 |
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Flat affect | 10016759 |
| Frustration tolerance decreased | 10077753 |
| Inappropriate affect | 10021588 |
| Irritability | 10022998 |
| Laziness | 10051602 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Moaning | 10027783 |
| Mood altered | 10027940 |
| Mood disorder due to a general medical condition | 10027944 |
| Mood swings | 10027951 |
| Morose | 10027977 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Premenstrual dysphoric disorder | 10051537 |
| Premenstrual syndrome | 10036618 |


| Screaming | 10039740 |
|---------------------------------|----------|
| Seasonal affective disorder | 10039775 |
| Steroid withdrawal syndrome | 10042028 |
| Substance-induced mood disorder | 10072387 |

### Anxiety

| PT | PT Code |
|-----------------------------------------------------|----------|
| Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10001084 |
| Aerophobia | 10080300 |
| Agitation | 10001497 |
| Agitation postoperative | 10049989 |
| Agoraphobia | 10001502 |
| Akathisia | 10001540 |
| Algophobia | 10078056 |
| Animal phobia | 10002518 |
| Anniversary reaction | 10074066 |
| Anticipatory anxiety | 10002758 |
| Anxiety | 10002855 |
| Anxiety disorder | 10057666 |
| Anxiety disorder due to a general medical condition | 10002859 |
| Arachnophobia | 10051408 |
| Astraphobia | 10078372 |
| Autophobia | 10071070 |
| Body dysmorphic disorder | 10052793 |
| Burnout syndrome | 10065369 |
| Catastrophic reaction | 10082329 |
| Cibophobia | 10082413 |
| Claustrophobia | 10009244 |
| Compulsions | 10010219 |
| Compulsive cheek biting | 10076510 |
| Compulsive handwashing | 10071263 |
| Compulsive hoarding | 10068007 |
| Compulsive lip biting | 10066241 |
| Compulsive shopping | 10067948 |
| Cryophobia | 10082662 |
| Dermatillomania | 10065701 |
| Dysmorphophobia | 10049096 |
| Emetophobia | 10070637 |
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |
| Fear of weight gain | 10016280 |
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |
| Haphephobia | 10067580 |


| Herpetophobia | 10081809 |
|---|---|
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosocomephobia | 10083993 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10003340 |
| Obsessive freed for symmetry Obsessive rumination | 10077179 |
| Obsessive furnification Obsessive thoughts | 10030204 |
| Obsessive trioughts Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive disorder Obsessive-compulsive symptom | 10029898 |
| Ochlophobia | 10077894 |
| Osmophobia | 10030093 |
| Paediatric autoimmune neuropsychiatric disorders associated with streptococcal infection | 10072147 |
| Panic attack | 10072147 |
| Panic disorder | 10033666 |
| Panic disorder Panic reaction | 10033670 |
| Paruresis | 10033670 |
| Performance fear | 10009024 |
| Phagophobia | 10054432 |
| Pharmacophobia | 10050096 |
| Phobia | 10009423 |
| Phobia of driving | 10054912 |
| Phobia of exams | 10036676 |
| Phobic avoidance | 10034918 |
| Phonophobia | 10054916 |
| Photaugiaphobia | 10034930 |
| Postpartum anxiety | 10082233 |
| Postpartum neurosis | 10082233 |
| Postpartum stress disorder | 10056394 |
| Post-traumatic stress disorder | 10036394 |
| Procedural anxiety | 10030310 |
| Pseudoangina | 10073204 |
| Selective mutism | 10030010 |
| Separation anxiety disorder | 10039917 |
| Sitophobia | 10040045 |
| Social anxiety disorder | 10080170 |
| Social fear | 10041247 |
| Stress | 10041247 |
| Tension | 10042209 |
| Terminal agitation | 10043208 |
| Thanatophobia | 10077410 |
| Thermophobia | 10004723 |
| Trichotemnomania | 10075147 |
| Trichotillomania | 10072732 |
| Hiorodillomania | 10044029 |

### **Sleep Disorders**

| PT | PT Code |
|------------------------------|----------|
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |


| Dehavioural induced insufficient aloon avadrams | 10081938 |
|---|---|
| Behavioural induced insufficient sleep syndrome Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Central-alveolar hypoventilation | 10007787 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Exploding head syndrome | 10080684 |
| Fatal familial insomnia | 10072077 |
| Hypersomnia | 10020765 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Insomnia related to another mental condition | 10022443 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Microsleep | 10076954 |
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Nightmare | 10029412 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Parasomnia | 10061910 |
| Paradoxical insomnia | 10083337 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep attacks | 10040981 |
| Sleep deficit | 10080881 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, parasomnia type | 10040988 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Somnolence | 10041349 |
| Somnolence neonatal | 10041350 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Sleep deficit | 10080881 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |


# Injection site Reactions Use CRF terms for ISR. Seizures/Convulsions

| PT | PT Code |
|-------------------------------------------------------------------|----------|
| 1p36 deletion syndrome | 10082398 |
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Alpers disease | 10083857 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| CEC syndrome | 10083749 |
| CDKL5 deficiency disorder | 10083005 |
| Change in seizure presentation | 10083003 |
| Clonic convulsion | 10073000 |
| Congenital bilateral perisylvian syndrome | 10033396 |
| Congenital bilateral pensylvian syndrome Convulsion in childhood | 10052391 |
| Convulsions local | 10032391 |
| Convulsive threshold lowered | 10010920 |
| CSWS syndrome | |
| | 10078827 |
| Deja vu | 10012177 |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst-suppression | 10071545 |
| Eclampsia | 10014129 |
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epilepsy with myoclonic-atonic seizures | 10081179 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Gelastic seizure | 10082918 |
| Generalised onset non-motor seizure | 10083376 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| GM2 gangliosidosis | 10083933 |
| Grey matter heterotopia | 10082084 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |
| Juvenile myoclonic epilepsy | 10071082 |
| Lafora's myoclonic epilepsy | 10071082 |
| Lennox-Gastaut syndrome | 10034030 |


| Migraine-triggered seizure | 10076676 |
|------------------------------------------------|----------|
| Molybdenum cofactor deficiency | 10069687 |
| Multiple subpial transection | 10079825 |
| Myoclonic epilepsy | 10054859 |
| Myoclonic epilepsy and ragged-red fibres | 10069825 |
| Neonatal epileptic seizure | 10082068 |
| Neonatal seizure | 10082067 |
| Partial seizures | 10061334 |
| Partial seizures with secondary generalisation | 10056209 |
| Petit mal epilepsy | 10034759 |
| Polymicrogyria | 10073489 |
| Post stroke epilepsy | 10076982 |
| Post stroke seizure | 10076981 |
| Postictal headache | 10052470 |
| Postictal paralysis | 10052469 |
| Postictal psychosis | 10070669 |
| Postictal state | 10048727 |
| Post-traumatic epilepsy | 10036312 |
| Schizencephaly | 10073487 |
| Seizure | 10039906 |
| Seizure anoxic | 10039907 |
| Seizure cluster | 10071350 |
| Seizure like phenomena | 10071048 |
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Transient epileptic amnesia | 10081728 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10050093 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

### Weight Gain

| PT | PT Code |
|-------------------------------|----------|
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |
| Weight abnormal | 10056814 |
| Weight increased | 10047899 |
| Waist circumference increased | 10064863 |
| Body mass index abnormal | 10074506 |
| Body mass index increased | 10005897 |
| Fat tissue increased | 10016251 |
| Sarcopenic obesity | 10083992 |

Rhabdomyolysis


| PT | PT Code |
|---------------------------|----------|
| Muscle necrosis | 10028320 |
| Myoglobin blood increased | 10028625 |
| Myoglobin blood present | 10059888 |
| Myoglobin urine present | 10028631 |
| Myoglobinaemia | 10058735 |
| Myoglobinuria | 10028629 |
| Myopathy | 10028641 |
| Myopathy toxic | 10028648 |
| Necrotising myositis | 10074769 |
| Rhabdomyolysis | 10039020 |
| Thyrotoxic myopathy | 10081524 |
| Myalgia | 10028411 |
| Myositis | 10028653 |

### **Pancreatitis**

| PT | PT Code |
|------------------------------------|----------|
| Cullen's sign | 10059029 |
| Grey Turner's sign | 10075426 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Hereditary pancreatitis | 10056976 |
| Immune-mediated pancreatitis | 10083072 |
| Ischaemic pancreatitis | 10066127 |
| Oedematous pancreatitis | 10052400 |
| Pancreatic abscess | 10048984 |
| Pancreatic cyst drainage | 10082531 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic necrosis | 10058096 |
| Pancreatic phlegmon | 10056975 |
| Pancreatic pseudoaneurysm | 10081762 |
| Pancreatic pseudocyst | 10033635 |
| Pancreatic pseudocyst drainage | 10033636 |
| Pancreatic pseudocyst haemorrhage | 10083813 |
| Pancreatic pseudocyst rupture | 10083811 |
| Pancreatitis | 10033645 |
| Pancreatitis acute | 10033647 |
| Pancreatitis haemorrhagic | 10033650 |
| Pancreatitis necrotising | 10033654 |
| Pancreatitis relapsing | 10033657 |
| Pancreatorenal syndrome | 10056277 |

**Impact on Creatinine** 

| PT | PT Code |
|-------------------------------|----------|
| Acute kidney injury | 10069339 |
| Acute phosphate nephropathy | 10069688 |
| Anuria | 10002847 |
| Azotaemia | 10003885 |
| Continuous haemodiafiltration | 10066338 |
| Dialysis | 10061105 |
| Foetal renal impairment | 10078987 |
| Haemodialysis | 10018875 |
| Haemofiltration | 10053090 |
| Neonatal anuria | 10049778 |
| Nephropathy toxic | 10029155 |
| Oliguria | 10030302 |
| Peritoneal dialysis | 10034660 |


| D 163 | 10070070 |
|--------------------------------------|----------|
| Prerenal failure | 10072370 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Atypical haemolytic uraemic syndrome | 10079840 |
| Cardiorenal syndrome | 10068230 |
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease | 10012660 |
| End stage renal disease | 10077512 |
| Haemolytic uraemic syndrome | 10018932 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Nail-patella syndrome | 10063431 |
| Pancreatorenal syndrome | 10056277 |
| Postoperative renal failure | 10056675 |
| Postrenal failure | 10059345 |
| Propofol infusion syndrome | 10063181 |
| Renal injury | 10061481 |
| Scleroderma renal crisis | 10062553 |
| Traumatic anuria | 10044501 |
